CLINICAL TRIAL: NCT05823974
Title: A Phase 1/2, Randomized, Dose-finding/Dose-confirmation Study to Evaluate the Reactogenicity, Safety and Immunogenicity of mRNA-based Multivalent Seasonal Influenza Vaccine Candidates Administered in Healthy Younger and Older Adults
Brief Title: A Study to Assess the Safety and Immune Response of a Vaccine Against Influenza in Healthy Younger and Older Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: CureVac (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 217884; 2022-502308-66-00 (Other: EU CT Number)
Record Dates: First submitted 2023-04-11; First posted 2023-04-21 (Actual); Results first posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-06

CONDITIONS: Influenza, Human
Keywords: Influenza; Safety; Reactogenicity; Immunogenicity; mRNA vaccine; Healthy younger adults; Healthy older adults
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Phase 2 of this study will be observer blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (21):
- Flu mRNA_Ph1_1 Younger Adults (YA) Group (Experimental): YA Participants received a single dose of Flu mRNA study intervention F2C22C/DL001Z (GSKVx000000039714) administered in Phase 1, at Day 1.
  Interventions: Biological: F2C22C/DL001Z
- Flu mRNA_Ph1_2 YA Group (Experimental): YA participants received a single dose of Flu mRNA study intervention F2B22A/DL001Z (GSKVx000000040038) administered in Phase 1, at Day 1.
  Interventions: Biological: F2B22A/DL001Z
- Flu mRNA_Ph1_3 YA Group (Experimental): YA participants received a single dose of Flu mRNA study intervention F2B22B/DL001Z (GSKVx000000040668) administered in Phase 1, at Day 1.
  Interventions: Biological: F2B22B/DL001Z
- Flu mRNA_Ph1_4 YA Group (Experimental): YA participants received a single dose of Flu mRNA study intervention F2B22C/DL001Z (GSKVx000000040671) administered in Phase 1, at Day 1.
  Interventions: Biological: F2B22C/DL001Z
- Flu mRNA_Ph1_5 YA Group (Experimental): YA participants received a single dose of Flu mRNA study intervention F2B22D/DL001Z (GSKVx000000040674) administered in Phase 1, at Day 1.
  Interventions: Biological: F2B22D/DL001Z
- Flu mRNA_Ph1_6 YA Group (Experimental): YA participants received a single dose of Flu mRNA study intervention F2B22E/DL001Z (GSKVx000000040677) administered in Phase 1, at Day 1.
  Interventions: Biological: F2B22E/DL001Z
- Flu mRNA_Ph1_7 YA Group (Experimental): YA participants received a single dose of Flu mRNA study intervention F2F22A/DL001Z (GSKVx000000040641) administered in Phase 1, at Day 1.
  Interventions: Biological: F2F22A/DL001Z
- Flu mRNA_Ph1_8 YA Group (Experimental): YA participants received a single dose of Flu mRNA study intervention F2F22B/DL001Z (GSKVx000000040644) administered in Phase 1, at Day 1.
  Interventions: Biological: F2F22B/DL001Z
- Flu mRNA_Ph1_9 YA Group (Experimental): YA participants received a single dose of Flu mRNA (GSK4382276A) study intervention F2F22C/DL001Z (GSKVx000000040647) administered in Phase 1, at Day 1.
  Interventions: Biological: F2F22C/DL001Z
- Flu mRNA_Ph1_10 YA Group (Experimental): YA participants received a single dose of Flu mRNA study intervention F2F22D/DL001Z (GSKVx000000040650) administered in Phase 1, at Day 1.
  Interventions: Biological: F2F22D/DL001Z
- Flu mRNA_Ph1_11 YA Group (Experimental): YA participants received a single dose of Flu mRNA study intervention F2F22E/DL001Z (GSKVx000000040996) administered in Phase 1, at Day 1.
  Interventions: Biological: F2F22E/DL001Z
- Flu mRNA_Ph1_12 YA Group (Experimental): YA participants received a single dose of Flu mRNA study intervention F2F22F/DL001Z (GSKVx000000040999) administered in Phase 1, at Day 1.
  Interventions: Biological: F2F22F/DL001Z
- Control Ph1_YA Group (Active Comparator): YA participants received a single dose of Control 1 administered in Phase 1, at Day 1.
  Interventions: Combination Product: Control 1
- Flu mRNA_Ph2_1_YA Group (Experimental): YA participants received a single dose of Flu mRNA study intervention F2F23D/DL001Z-NH administered in Phase 2, at Day 1.
  Interventions: Biological: F2F23D/DL001Z-NH
- Flu mRNA_Ph2_2_YA Group (Experimental): YA participants received a single dose of Flu mRNA study intervention F2F23A/DL001Z-NH administered in Phase 2, at Day 1.
  Interventions: Biological: F2F23A/DL001Z-NH
- Flu mRNA_Ph2_3_YA Group (Experimental): YA participants received a single dose of Flu mRNA study intervention F2F23B/DL001Z-NH administered in Phase 2, at Day 1.
  Interventions: Biological: F2F23B/DL001Z-NH
- Control_Ph2_YA Group (Active Comparator): YA participants received single dose of Control 2 vaccine administered in Phase 2, at Day 1.
  Interventions: Combination Product: Control 2
- Flu mRNA_Ph2_1_Older adults (OA) Group (Experimental): OA participants received a single dose of Flu mRNA study intervention F2F23A/DL001Z-NH administered in Phase 2, at Day 1.
  Interventions: Biological: F2F23A/DL001Z-NH
- Flu mRNA_Ph2_2_OA Group (Experimental): OA participants received a single dose of Flu mRNA study intervention F2F23B/DL001Z-NH administered in Phase 2, at Day 1.
  Interventions: Biological: F2F23B/DL001Z-NH
- Flu mRNA_Ph2_3_OA Group (Experimental): OA participants received a single dose of Flu mRNA study intervention F2F23C/DL001Z-NH administered in Phase 2, at Day 1.
  Interventions: Biological: F2F23C/DL001Z-NH
- Control_Ph2_OA Group (Active Comparator): OA participants received a single dose of Control 3 vaccine administered in Phase 2, at Day 1.
  Interventions: Combination Product: Control 3

INTERVENTIONS:
Biological: F2C22C/DL001Z — Study intervention was administered intramuscularly in Phase 1, at Day 1.
  Arms: Flu mRNA_Ph1_1 Younger Adults (YA) Group
Biological: F2B22A/DL001Z — Study intervention was administered intramuscularly in Phase 1, at Day 1.
  Arms: Flu mRNA_Ph1_2 YA Group
Biological: F2B22B/DL001Z — Study intervention was administered intramuscularly in Phase 1, at Day 1.
  Arms: Flu mRNA_Ph1_3 YA Group
Biological: F2B22C/DL001Z — Study intervention was administered intramuscularly in Phase 1, at Day 1.
  Arms: Flu mRNA_Ph1_4 YA Group
Biological: F2B22D/DL001Z — Study intervention was administered intramuscularly in Phase 1, at Day 1.
  Arms: Flu mRNA_Ph1_5 YA Group
Biological: F2B22E/DL001Z — Study intervention was administered intramuscularly in Phase 1, at Day 1.
  Arms: Flu mRNA_Ph1_6 YA Group
Biological: F2F22A/DL001Z — Study intervention was administered intramuscularly in Phase 1, at Day 1.
  Arms: Flu mRNA_Ph1_7 YA Group
Biological: F2F22B/DL001Z — Study intervention was administered intramuscularly in Phase 1, at Day 1.
  Arms: Flu mRNA_Ph1_8 YA Group
Biological: F2F22C/DL001Z — Study intervention was administered intramuscularly in Phase 1, at Day 1.
  Arms: Flu mRNA_Ph1_9 YA Group
Biological: F2F22D/DL001Z — Study intervention was administered intramuscularly in Phase 1, at Day 1.
  Arms: Flu mRNA_Ph1_10 YA Group
Biological: F2F22E/DL001Z — Study intervention was administered intramuscularly in Phase 1, at Day 1.
  Arms: Flu mRNA_Ph1_11 YA Group
Combination Product: Control 1 — Control vaccine was administered intramuscularly in Phase 1, at Day 1.
  Arms: Control Ph1_YA Group
Biological: F2F23D/DL001Z-NH — Study intervention was administered intramuscularly in Phase 2, at Day 1.
  Arms: Flu mRNA_Ph2_1_YA Group
Biological: F2F23A/DL001Z-NH — Study intervention was administered intramuscularly in Phase 2, at Day 1.
  Arms: Flu mRNA_Ph2_1_Older adults (OA) Group; Flu mRNA_Ph2_2_YA Group
Biological: F2F23B/DL001Z-NH — Study intervention was administered intramuscularly in Phase 2, at Day 1.
  Arms: Flu mRNA_Ph2_2_OA Group; Flu mRNA_Ph2_3_YA Group
Combination Product: Control 2 — Control vaccine was administered intramuscularly in Phase 2, at Day 1.
  Arms: Control_Ph2_YA Group
Biological: F2F23C/DL001Z-NH — Study intervention was administered intramuscularly in Phase 2, at Day 1.
  Arms: Flu mRNA_Ph2_3_OA Group
Combination Product: Control 3 — Control vaccine was administered intramuscularly in Phase 2, at Day 1.
  Arms: Control_Ph2_OA Group
Biological: F2F22F/DL001Z — Study intervention was administered intramuscularly in Phase 1, at Day 1.
  Arms: Flu mRNA_Ph1_12 YA Group

SUMMARY:
The purpose of this study is to find and confirm the dose and asses the reactogenicity, safety and immune response of GlaxoSmithKline's (GSK) messenger RNA (mRNA)-based multivalent seasonal influenza vaccine (GSK4382276A) candidates administered in healthy younger and older adults (OA).

ELIGIBILITY:
Inclusion Criteria:

* A male or female between and including 18 and 50 years of age in Phase 1 and between and including 18 and 85 years of age (YA: 18-64; OA: 65-85) in Phase 2 at the time of the study intervention administration.
* Healthy participants or medically stable participants as established by medical history, clinical examination, and safety laboratory assessments. Participants with chronic medical conditions with or without specific treatment are allowed to participate in this study if considered by the investigator as medically stable. A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization for worsening disease during 3 months before enrollment.
* Body mass index (BMI) >=18 kilograms per meter square (kg/m^2) and less than or equal to (<=) 35 kg/m^2.
* Participants who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent obtained from the participant prior to performing any study-specific procedure.
* Female participants of non-childbearing potential may be enrolled in the study.
* Female participants of childbearing potential may be enrolled in the study if the participant:
* has practiced adequate contraception for 28 days prior to study intervention administration, and
* has a negative pregnancy test on the day of study intervention administration, and
* has agreed to continue adequate contraception for at least 1 month after study intervention administration

Exclusion Criteria:

Medical conditions

* Only in Phase 1: Any clinically significant* hematological, biochemical, urinalysis or (hemoglobin A1c) HbA1c laboratory abnormality.

  *The investigator should use the clinical judgment to decide which abnormalities are clinically significant.
* Participant tested positive for influenza by local health authority-approved testing methods within 180 days prior to Day 1.
* Current or past malignancy, unless completely resolved without clinically significant sequelae for >5 years.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including HIV infection, based on medical history and physical examination (no laboratory testing required). However, in Phase 2, HIV-infected individuals may be enrolled if participants have been stable on antiretroviral therapy for the past 6 consecutive months, i.e., their treatment has not been modified, their cluster of differentiation 4 (CD4) cell count is >=200/cubic millimeter (mm^3) and their viral load has been undetectable (i.e., HIV-RNA less than (<) 50 copies/milliliter [mL]) (based on medical records, no laboratory testing required).
* History of myocarditis or pericarditis less than or equal to 10 years prior to vaccine administration, including a history of myocarditis or pericarditis following vaccination with an mRNA coronavirus disease 2019 (COVID-19) vaccine.
* Participants with history of hypersensitivity or severe allergic reaction to any previous vaccine or hypersensitivity likely to be exacerbated by any component of the study intervention (including latex, polyethylene glycol, egg protein and aminoglycoside antibiotics).
* History of, or uncontrolled neurological disorders or seizures, including Guillain-Barré syndrome and Bell's palsy, with the exception of febrile seizures during childhood.
* Any history of dementia or any medical condition that moderately or severely impairs cognition.
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.

Prior/Concomitant therapy

* Administration of an influenza vaccine (including any of the study investigational vaccines) within 180 days before enrollment or planned administration within 28 days (Day 29) after the study intervention administration.
* Phase 1: Administration of a vaccine not foreseen by the study protocol in the period starting 28 days (Day -28) before the study intervention administration or planned administration within 28 days (Day 29) after the study intervention administration. Phase 2: Administration of a vaccine not foreseen by the study protocol in the period starting 15 days (Day -15) before the study intervention administration or planned administration within 28 days (Day 29) after the study intervention administration.

  *In case emergency mass vaccination for an unforeseen public health threat is recommended and/or organized by public health authorities outside the routine immunization program, the time period described above can be reduced to 7 days if, necessary for that vaccine, provided it is used according to the local governmental recommendations and that the Sponsor is notified accordingly.
* Use of any investigational or non-registered product (drug, vaccine, or invasive medical device) other than the study intervention during the period beginning 30 days before the study intervention administration, or their planned use during the study period.
* Administration of long-acting immune-modifying drugs within 90 days before enrollment or planned use at any time during the study period.
* Administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 90 days before the study intervention administration, or planned administration during the study period. Administration of monoclonal antibodies specifically directed against the spike protein of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2), for treatment of COVID-19 disease is allowed.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting 3 months prior to the study intervention administration. For corticosteroids, this will mean prednisone equivalent >=20 milligrams (mg)/day. Inhaled, topical and intraarticular steroids are allowed.

Other exclusions

* Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational intervention (drug/invasive medical device).
* Pregnant or lactating female.
* Bedridden participants.
* Female planning to become pregnant or planning to discontinue contraceptive precautions within the 1-month post-dosing period.
* Alcoholism or substance use disorder within the past 24 months based on the presence of 2 or more of the following abuse criteria: hazardous use, social/interpersonal problems related to use, neglect of major roles to use, withdrawal, tolerance, use of larger amounts or longer, repeated attempts to quit or control use, much time spent using, physical or psychological problems related to use, activities given up to use, craving.
* Any study personnel or their immediate dependents, family, or household members.
* Participants with extensive tattoos covering deltoid region on both arms that would preclude the assessment of local reactogenicity.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1275 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (41):
- United States (24):
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Valparaiso, Indiana
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Dearborn, Michigan
  - GSK Investigational Site, Papillion, Nebraska
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Denver, North Carolina
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, East Greenwich, Rhode Island
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Tomball, Texas
  - GSK Investigational Site, Newport News, Virginia
  - GSK Investigational Site, Norfolk, Virginia
- Belgium (8):
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Ieper
  - GSK Investigational Site, Kluisbergen
  - GSK Investigational Site, Mechelen
  - GSK Investigational Site, Tielt
  - GSK Investigational Site, Zwalm
- Canada (5):
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Chicoutimi, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- South Africa (4):
  - GSK Investigational Site, Buffalo
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Johannesburg
  - GSK Investigational Site, Tembisa

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1275 participants were included in Enrolled set, out of which only 1256 were included in Exposed set and started the study.
Period: Overall Study
Arm/Group | Flu mRNA_Ph1_1 Younger Adults (YA) Group | Flu mRNA_Ph1_2 YA Group | Flu mRNA_Ph1_3 YA Group | Flu mRNA_Ph1_4 YA Group | Flu mRNA_Ph1_5 YA Group | Flu mRNA_Ph1_6 YA Group | Flu mRNA_Ph1_7 YA Group | Flu mRNA_Ph1_8 YA Group | Flu mRNA_Ph1_9 YA Group | Flu mRNA_Ph1_10 YA Group | Flu mRNA_Ph1_11 YA Group | Flu mRNA_Ph1_12 YA Group | Control Ph1_YA Group | Flu mRNA_Ph2_1_YA Group | Flu mRNA_Ph2_2_YA Group | Flu mRNA_Ph2_3_YA Group | Control_Ph2_YA Group | Flu mRNA_Ph2_1_Older Adults (OA) Group | Flu mRNA_Ph2_2_OA Group | Flu mRNA_Ph2_3_OA Group | Control_Ph2_OA Group
Started | 21 | 22 | 23 | 23 | 22 | 25 | 23 | 22 | 23 | 22 | 23 | 21 | 23 | 115 | 108 | 137 | 120 | 119 | 122 | 125 | 117
Completed | 20 | 17 | 18 | 22 | 19 | 21 | 20 | 20 | 20 | 20 | 21 | 21 | 20 | 111 | 105 | 131 | 119 | 116 | 119 | 123 | 116
Not Completed | 1 | 5 | 5 | 1 | 3 | 4 | 3 | 2 | 3 | 2 | 2 | 0 | 3 | 4 | 3 | 6 | 1 | 3 | 3 | 2 | 1
Not completed — Lost to Follow-up | 0 | 3 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 2 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 2 | 0 | 2 | 3 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 1 | 3 | 0 | 2 | 2 | 0 | 1
Not completed — MIGRATED / MOVED FROM THE STUDY AREA | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Flu mRNA_Ph1_1 Younger Adults (YA) Group | Flu mRNA_Ph1_2 YA Group | Flu mRNA_Ph1_3 YA Group | Flu mRNA_Ph1_4 YA Group | Flu mRNA_Ph1_5 YA Group | Flu mRNA_Ph1_6 YA Group | Flu mRNA_Ph1_7 YA Group | Flu mRNA_Ph1_8 YA Group | Flu mRNA_Ph1_9 YA Group | Flu mRNA_Ph1_10 YA Group | Flu mRNA_Ph1_11 YA Group | Flu mRNA_Ph1_12 YA Group | Control Ph1_YA Group | Flu mRNA_Ph2_1_YA Group | Flu mRNA_Ph2_2_YA Group | Flu mRNA_Ph2_3_YA Group | Control_Ph2_YA Group | Flu mRNA_Ph2_1_Older Adults (OA) Group | Flu mRNA_Ph2_2_OA Group | Flu mRNA_Ph2_3_OA Group | Control_Ph2_OA Group | Total
Number analyzed (Participants) | 21 | 22 | 23 | 23 | 22 | 25 | 23 | 22 | 23 | 22 | 23 | 21 | 23 | 115 | 108 | 137 | 120 | 119 | 122 | 125 | 117 | 1256
Age, Customized [Count of Participants; unit: Participants]
  18 - 64 years | 21 | 22 | 23 | 23 | 22 | 25 | 23 | 22 | 23 | 22 | 23 | 21 | 23 | 114 | 108 | 137 | 120 | 1 | 0 | 0 | 0 | 773
  65 - 84 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 118 | 121 | 124 | 117 | 481
  ≥ 85 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 15 | 13 | 13 | 13 | 11 | 13 | 13 | 11 | 12 | 13 | 8 | 65 | 55 | 86 | 70 | 69 | 55 | 61 | 71 | 690
  Male | 9 | 11 | 8 | 10 | 9 | 12 | 12 | 9 | 10 | 11 | 11 | 8 | 15 | 50 | 53 | 51 | 50 | 50 | 67 | 64 | 46 | 566
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — The "All Other Races" category (i.e., American Indian or Alaska Native, Asian and Black or African American for phase 1 YA and phase II YA & OA, where 0<n<11) are combined into one category to maintain participant confidentiality and privacy.
  Participants
    WHITE | 14 | 19 | 19 | 18 | 16 | 18 | 16 | 19 | 17 | 15 | 17 | 13 | 19 | 94 | 91 | 116 | 96 | 88 | 95 | 101 | 87 | 988
    All other Races | 5 | 2 | 4 | 5 | 6 | 6 | 7 | 3 | 6 | 7 | 6 | 8 | 4 | 19 | 15 | 19 | 17 | 25 | 22 | 19 | 21 | 226
    MULTIPLE | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 1 | 0 | 1 | 9
    NOT REPORTED | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 3 | 5 | 4 | 5 | 8 | 31
    UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Any Solicited Administration Site Adverse Events (AEs)
Description: Assessed solicited administration site events included pain, redness (Erythema), swelling, lymphadenopathy (defined as localized axillary, cervical or supraclavicular swelling or tenderness ipsilateral to the injection arm). Any = occurrence of the event regardless of intensity grade or relation to the study vaccination.
Time Frame: Day 1 to Day 7
Population: The analysis was performed on the Exposed Set (ES), which included all participants who received a study intervention and for whom solicited administration site events data were available at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Flu mRNA_Ph1_1 Younger Adults (YA) Group | Flu mRNA_Ph1_2 YA Group | Flu mRNA_Ph1_3 YA Group | Flu mRNA_Ph1_4 YA Group | Flu mRNA_Ph1_5 YA Group | Flu mRNA_Ph1_6 YA Group | Flu mRNA_Ph1_7 YA Group | Flu mRNA_Ph1_8 YA Group | Flu mRNA_Ph1_9 YA Group | Flu mRNA_Ph1_10 YA Group | Flu mRNA_Ph1_11 YA Group | Flu mRNA_Ph1_12 YA Group | Control Ph1_YA Group | Flu mRNA_Ph2_1_YA Group | Flu mRNA_Ph2_2_YA Group | Flu mRNA_Ph2_3_YA Group | Control_Ph2_YA Group | Flu mRNA_Ph2_1_Older Adults (OA) Group | Flu mRNA_Ph2_2_OA Group | Flu mRNA_Ph2_3_OA Group | Control_Ph2_OA Group
Number analyzed (Participants) | 21 | 22 | 23 | 23 | 22 | 25 | 23 | 21 | 23 | 22 | 23 | 21 | 23 | 115 | 108 | 137 | 120 | 119 | 122 | 125 | 117
Participants
  Erythema | 0 | 2 | 2 | 2 | 3 | 4 | 1 | 1 | 1 | 3 | 3 | 3 | 2 | 3 | 5 | 8 | 1 | 6 | 6 | 9 | 4
  Lymphadenopathy | 6 | 10 | 8 | 10 | 10 | 14 | 5 | 9 | 8 | 10 | 8 | 11 | 2 | 28 | 41 | 53 | 14 | 20 | 19 | 14 | 10
  Pain | 15 | 19 | 21 | 20 | 19 | 22 | 15 | 19 | 18 | 19 | 21 | 18 | 13 | 82 | 86 | 118 | 53 | 63 | 64 | 78 | 41
  Swelling | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 2 | 3 | 0 | 3 | 3 | 2 | 3 | 7 | 7 | 1 | 6 | 5 | 8 | 6

2. Primary Outcome: Number of Participants Reporting Any Solicited Systemic AEs
Description: Assessed solicited systemic events included fever (defined as axillary temperature greater than or equal to (>=) 38.0°C/100.4°F), chills, headache, fatigue, myalgia, and arthralgia. Any = occurrence of the event regardless of intensity grade or relation to the study vaccination.
Time Frame: Day 1 to Day 7
Population: The analysis was performed on the ES, which included all participants who received a study intervention and for whom solicited systemic events data were available at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Flu mRNA_Ph1_1 Younger Adults (YA) Group | Flu mRNA_Ph1_2 YA Group | Flu mRNA_Ph1_3 YA Group | Flu mRNA_Ph1_4 YA Group | Flu mRNA_Ph1_5 YA Group | Flu mRNA_Ph1_6 YA Group | Flu mRNA_Ph1_7 YA Group | Flu mRNA_Ph1_8 YA Group | Flu mRNA_Ph1_9 YA Group | Flu mRNA_Ph1_10 YA Group | Flu mRNA_Ph1_11 YA Group | Flu mRNA_Ph1_12 YA Group | Control Ph1_YA Group | Flu mRNA_Ph2_1_YA Group | Flu mRNA_Ph2_2_YA Group | Flu mRNA_Ph2_3_YA Group | Control_Ph2_YA Group | Flu mRNA_Ph2_1_Older Adults (OA) Group | Flu mRNA_Ph2_2_OA Group | Flu mRNA_Ph2_3_OA Group | Control_Ph2_OA Group
Number analyzed (Participants) | 21 | 22 | 23 | 23 | 22 | 25 | 23 | 21 | 23 | 22 | 23 | 21 | 23 | 115 | 108 | 137 | 120 | 119 | 122 | 125 | 117
Participants
  Arthralgia | 3 | 12 | 8 | 10 | 11 | 10 | 9 | 11 | 11 | 7 | 9 | 10 | 0 | 31 | 37 | 48 | 11 | 15 | 27 | 33 | 9
  Chills | 4 | 12 | 11 | 14 | 10 | 9 | 15 | 15 | 12 | 12 | 20 | 13 | 0 | 30 | 39 | 73 | 18 | 18 | 19 | 37 | 7
  Fatigue | 10 | 19 | 17 | 18 | 17 | 18 | 16 | 19 | 17 | 16 | 18 | 17 | 9 | 58 | 70 | 103 | 49 | 44 | 51 | 64 | 26
  Headache | 11 | 17 | 15 | 17 | 16 | 17 | 15 | 17 | 14 | 16 | 17 | 13 | 5 | 54 | 58 | 99 | 36 | 36 | 36 | 50 | 19
  Myalgia | 10 | 21 | 15 | 18 | 15 | 19 | 15 | 16 | 16 | 18 | 20 | 18 | 9 | 56 | 70 | 98 | 35 | 36 | 40 | 57 | 19
  Temperature | 1 | 2 | 6 | 10 | 4 | 1 | 8 | 5 | 7 | 5 | 9 | 6 | 0 | 5 | 8 | 25 | 2 | 1 | 5 | 14 | 2

3. Primary Outcome: Number of Participants Reporting Any Unsolicited AEs
Description: An unsolicited AE is defined as an AE that was either not included in the list of solicited events or could be included in the list of solicited events but with an onset outside the specified period of follow up for solicited events. Unsolicited AEs include both serious and non-serious AEs. Any = occurrence the event regardless of intensity grade or relation to the study vaccination.
Time Frame: Day 1 to Day 28
Population: The analysis was performed on the ES, which included all participants who received a study intervention and for whom unsolicited AEs data were available at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Flu mRNA_Ph1_1 Younger Adults (YA) Group | Flu mRNA_Ph1_2 YA Group | Flu mRNA_Ph1_3 YA Group | Flu mRNA_Ph1_4 YA Group | Flu mRNA_Ph1_5 YA Group | Flu mRNA_Ph1_6 YA Group | Flu mRNA_Ph1_7 YA Group | Flu mRNA_Ph1_8 YA Group | Flu mRNA_Ph1_9 YA Group | Flu mRNA_Ph1_10 YA Group | Flu mRNA_Ph1_11 YA Group | Flu mRNA_Ph1_12 YA Group | Control Ph1_YA Group | Flu mRNA_Ph2_1_YA Group | Flu mRNA_Ph2_2_YA Group | Flu mRNA_Ph2_3_YA Group | Control_Ph2_YA Group | Flu mRNA_Ph2_1_Older Adults (OA) Group | Flu mRNA_Ph2_2_OA Group | Flu mRNA_Ph2_3_OA Group | Control_Ph2_OA Group
Number analyzed (Participants) | 21 | 22 | 23 | 23 | 22 | 25 | 23 | 22 | 23 | 22 | 23 | 21 | 23 | 115 | 108 | 137 | 120 | 119 | 122 | 125 | 117
Participants | 7 | 10 | 5 | 7 | 6 | 12 | 4 | 6 | 12 | 8 | 7 | 9 | 7 | 34 | 40 | 60 | 45 | 24 | 22 | 28 | 20

4. Primary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs)
Description: An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant, is an abnormal pregnancy outcome, or is a suspected transmission of any infectious agent via an authorized medicinal product. Any = occurrence the event regardless of intensity grade or relation to the study vaccination.
Time Frame: Day 1 to Day 183
Population: The analysis was performed on the ES, which included all participants who received a study intervention and for whom SAEs data were available at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Flu mRNA_Ph1_1 Younger Adults (YA) Group | Flu mRNA_Ph1_2 YA Group | Flu mRNA_Ph1_3 YA Group | Flu mRNA_Ph1_4 YA Group | Flu mRNA_Ph1_5 YA Group | Flu mRNA_Ph1_6 YA Group | Flu mRNA_Ph1_7 YA Group | Flu mRNA_Ph1_8 YA Group | Flu mRNA_Ph1_9 YA Group | Flu mRNA_Ph1_10 YA Group | Flu mRNA_Ph1_11 YA Group | Flu mRNA_Ph1_12 YA Group | Control Ph1_YA Group | Flu mRNA_Ph2_1_YA Group | Flu mRNA_Ph2_2_YA Group | Flu mRNA_Ph2_3_YA Group | Control_Ph2_YA Group | Flu mRNA_Ph2_1_Older Adults (OA) Group | Flu mRNA_Ph2_2_OA Group | Flu mRNA_Ph2_3_OA Group | Control_Ph2_OA Group
Number analyzed (Participants) | 21 | 22 | 23 | 23 | 22 | 25 | 23 | 22 | 23 | 22 | 23 | 21 | 23 | 115 | 108 | 137 | 120 | 119 | 122 | 125 | 117
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 3 | 6 | 2 | 2

5. Primary Outcome: Number of Participants Reporting AEs of Special Interest (AESIs)
Description: The following events were considered as AESI in this study: severe hypersensitivity reactions within 24 hours after study intervention administration, myocarditis/pericarditis and potential immune-mediated diseases (pIMDs). Any = occurrence the event regardless of intensity grade or relation to the study vaccination.
Time Frame: Day 1 to Day 183
Population: The analysis was performed on the ES, which included all participants who received a study intervention and for whom AESI data were available at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Flu mRNA_Ph1_1 Younger Adults (YA) Group | Flu mRNA_Ph1_2 YA Group | Flu mRNA_Ph1_3 YA Group | Flu mRNA_Ph1_4 YA Group | Flu mRNA_Ph1_5 YA Group | Flu mRNA_Ph1_6 YA Group | Flu mRNA_Ph1_7 YA Group | Flu mRNA_Ph1_8 YA Group | Flu mRNA_Ph1_9 YA Group | Flu mRNA_Ph1_10 YA Group | Flu mRNA_Ph1_11 YA Group | Flu mRNA_Ph1_12 YA Group | Control Ph1_YA Group | Flu mRNA_Ph2_1_YA Group | Flu mRNA_Ph2_2_YA Group | Flu mRNA_Ph2_3_YA Group | Control_Ph2_YA Group | Flu mRNA_Ph2_1_Older Adults (OA) Group | Flu mRNA_Ph2_2_OA Group | Flu mRNA_Ph2_3_OA Group | Control_Ph2_OA Group
Number analyzed (Participants) | 21 | 22 | 23 | 23 | 22 | 25 | 23 | 22 | 23 | 22 | 23 | 21 | 23 | 115 | 108 | 137 | 120 | 119 | 122 | 125 | 117
Participants | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0

6. Primary Outcome: Number of Participants Reporting Medically Attended Events (MAEs)
Description: MAE is defined as an AE that results in an unscheduled visit to a medical professional (e.g., physician's office visits, emergency room visits or hospitalization). Any = occurrence the event regardless of intensity grade or relation to the study vaccination.
Time Frame: Day 1 to Day 183
Population: The analysis was performed on the ES, which included all participants who received a study intervention and for whom MAEs data were available at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Flu mRNA_Ph1_1 Younger Adults (YA) Group | Flu mRNA_Ph1_2 YA Group | Flu mRNA_Ph1_3 YA Group | Flu mRNA_Ph1_4 YA Group | Flu mRNA_Ph1_5 YA Group | Flu mRNA_Ph1_6 YA Group | Flu mRNA_Ph1_7 YA Group | Flu mRNA_Ph1_8 YA Group | Flu mRNA_Ph1_9 YA Group | Flu mRNA_Ph1_10 YA Group | Flu mRNA_Ph1_11 YA Group | Flu mRNA_Ph1_12 YA Group | Control Ph1_YA Group | Flu mRNA_Ph2_1_YA Group | Flu mRNA_Ph2_2_YA Group | Flu mRNA_Ph2_3_YA Group | Control_Ph2_YA Group | Flu mRNA_Ph2_1_Older Adults (OA) Group | Flu mRNA_Ph2_2_OA Group | Flu mRNA_Ph2_3_OA Group | Control_Ph2_OA Group
Number analyzed (Participants) | 21 | 22 | 23 | 23 | 22 | 25 | 23 | 22 | 23 | 22 | 23 | 21 | 23 | 115 | 108 | 137 | 120 | 119 | 122 | 125 | 117
Participants | 3 | 3 | 4 | 3 | 2 | 7 | 3 | 3 | 3 | 3 | 2 | 8 | 6 | 28 | 28 | 29 | 30 | 20 | 21 | 17 | 18

7. Primary Outcome: Number of Participants Reporting a Shift From Abnormal Non-clinically Significant and Normal or Missing Laboratory Value on Day 1 to Clinically Significant Abnormal Laboratory Value on Day 8 for Hematology, and Clinical Chemistry
Description: Clinically significant abnormal laboratory findings are those which are not associated with an underlying disease, unless judged by the investigator to be more severe than expected for the participants condition. Normal or missing values refer to laboratory values that were within normal range or missing at baseline.
Time Frame: At Day 8 compared to baseline (Day 1)
Population: The analysis was performed on the ES, which included all participants who received a study intervention and for whom laboratory data were available at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Flu mRNA_Ph1_1 Younger Adults (YA) Group | Flu mRNA_Ph1_2 YA Group | Flu mRNA_Ph1_3 YA Group | Flu mRNA_Ph1_4 YA Group | Flu mRNA_Ph1_5 YA Group | Flu mRNA_Ph1_6 YA Group | Flu mRNA_Ph1_7 YA Group | Flu mRNA_Ph1_8 YA Group | Flu mRNA_Ph1_9 YA Group | Flu mRNA_Ph1_10 YA Group | Flu mRNA_Ph1_11 YA Group | Flu mRNA_Ph1_12 YA Group | Control Ph1_YA Group
Number analyzed (Participants) | 21 | 22 | 23 | 23 | 21 | 25 | 23 | 22 | 23 | 21 | 23 | 21 | 23
Participants
  Abnormal non-significant to clinically significant | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Normal or missing to clinically significant | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 2 | 1 | 0 | 0 | 1

8. Primary Outcome: Number of Participants Reporting a Shift From Abnormal Non-clinically Significant and Normal or Missing Laboratory Value on Day 1 to Clinically Significant Abnormal Laboratory Value on Day 29 for Hematology, and Clinical Chemistry
Description: as for outcome 7
Time Frame: At Day 29 compared to baseline (Day 1)
Population: The analysis was performed on the ES, which included all participants who received a study intervention and for whom laboratory data were available for the specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Flu mRNA_Ph1_1 Younger Adults (YA) Group | Flu mRNA_Ph1_2 YA Group | Flu mRNA_Ph1_3 YA Group | Flu mRNA_Ph1_4 YA Group | Flu mRNA_Ph1_5 YA Group | Flu mRNA_Ph1_6 YA Group | Flu mRNA_Ph1_7 YA Group | Flu mRNA_Ph1_8 YA Group | Flu mRNA_Ph1_9 YA Group | Flu mRNA_Ph1_10 YA Group | Flu mRNA_Ph1_11 YA Group | Flu mRNA_Ph1_12 YA Group | Control Ph1_YA Group
Number analyzed (Participants) | 20 | 22 | 22 | 23 | 21 | 25 | 23 | 22 | 21 | 21 | 22 | 21 | 22
Participants
  Abnormal non-significant to clinically significant | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Normal or missing to clinically significant | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Geometric Mean Titer (GMT) of Antigen 1 Antibody Titer
Description: Assay 1= with egg propagated Influenza virus and Assay 2= with cell propagated Influenza virus.
Time Frame: At Day 29
Population: The analysis was performed on the Per Protocol Set (PPS), which included all eligible participants who received the study intervention dose according to the protocol, had recorded anti-HI immunogenicity results pre- and post-dose, without intercurrent conditions, and did not use prohibited medications or vaccinations before Day 29 and for whom data were available for the specified analysis at the specified timepoints. Blood sample results that deviated from the analysis criteria were excluded.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Flu mRNA_Ph1_1 Younger Adults (YA) Group | Flu mRNA_Ph1_2 YA Group | Flu mRNA_Ph1_3 YA Group | Flu mRNA_Ph1_4 YA Group | Flu mRNA_Ph1_5 YA Group | Flu mRNA_Ph1_6 YA Group | Flu mRNA_Ph1_7 YA Group | Flu mRNA_Ph1_8 YA Group | Flu mRNA_Ph1_9 YA Group | Flu mRNA_Ph1_10 YA Group | Flu mRNA_Ph1_11 YA Group | Flu mRNA_Ph1_12 YA Group | Control Ph1_YA Group | Flu mRNA_Ph2_1_YA Group | Flu mRNA_Ph2_2_YA Group | Flu mRNA_Ph2_3_YA Group | Control_Ph2_YA Group | Flu mRNA_Ph2_1_Older Adults (OA) Group | Flu mRNA_Ph2_2_OA Group | Flu mRNA_Ph2_3_OA Group | Control_Ph2_OA Group
Number analyzed (Participants) | 19 | 22 | 22 | 23 | 21 | 24 | 23 | 22 | 19 | 21 | 22 | 19 | 22 | 101 | 97 | 121 | 115 | 108 | 116 | 115 | 111
Titers
  Flu A1 Assay 1: number analyzed (Participants) | 19 | 22 | 22 | 23 | 21 | 24 | 23 | 22 | 19 | 21 | 22 | 19 | 22 | 101 | 94 | 119 | 114 | 107 | 112 | 113 | 111
  Flu A1 Assay 1 | 469.49 [300.51 to 733.47] | 335.19 [222.96 to 503.91] | 247.82 [164.81 to 372.65] | 359.26 [240.96 to 535.62] | 380.39 [249.53 to 579.90] | 331.81 [224.48 to 490.45] | 349.06 [233.45 to 521.94] | 324.35 [215.04 to 489.23] | 409.93 [264.86 to 634.45] | 370.39 [243.46 to 563.51] | 308.20 [204.25 to 465.06] | 341.20 [219.93 to 529.33] | 224.76 [148.16 to 340.98] | 50.99 [40.14 to 64.76] | 62.65 [49.16 to 79.83] | 75.46 [60.58 to 94.01] | 46.97 [37.55 to 58.75] | 59.83 [46.90 to 76.33] | 81.06 [63.87 to 102.88] | 90.00 [70.89 to 114.26] | 56.52 [44.51 to 71.77]
  Flu A1 Assay 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 0 | 0 | 0 | 0 | 0 | 0 | 101 | 97 | 121 | 114 | 108 | 115 | 115 | 111
  Flu A1 Assay 2 |  |  |  |  |  |  | 103.70 [64.91 to 165.68] |  |  |  |  |  |  | 262.86 [209.06 to 330.49] | 260.70 [207.26 to 327.92] | 292.27 [237.21 to 360.11] | 175.58 [141.75 to 217.49] | 255.17 [202.02 to 322.31] | 287.14 [228.87 to 360.24] | 338.20 [269.10 to 425.06] | 176.21 [139.85 to 222.01]
  Flu A2 Assay 1 | 15.64 [10.04 to 24.38] | 135.68 [90.45 to 203.53] | 90.47 [60.32 to 135.69] | 143.63 [96.56 to 213.64] | 87.87 [57.78 to 133.64] | 98.27 [66.61 to 144.97] | 87.80 [58.95 to 130.79] | 97.63 [64.85 to 146.98] | 110.15 [71.25 to 170.27] | 99.75 [65.65 to 151.56] | 135.41 [90.11 to 203.47] | 88.55 [57.18 to 137.14] | 38.02 [25.13 to 57.52] | 98.57 [79.34 to 122.45] | 113.45 [91.29 to 141.00] | 143.74 [117.88 to 175.28] | 58.80 [48.00 to 72.02] | 159.66 [127.81 to 199.45] | 160.93 [129.62 to 199.79] | 191.29 [153.92 to 237.74] | 107.50 [86.28 to 133.94]
  Flu A2 Assay 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 0 | 19 | 0 | 0 | 0 | 0 | 101 | 97 | 121 | 114 | 108 | 115 | 115 | 111
  Flu A2 Assay 2 |  |  |  |  |  |  | 295.42 [182.26 to 478.85] |  | 1545.64 [921.87 to 2591.47] |  |  |  |  | 436.01 [347.19 to 547.55] | 469.09 [373.13 to 589.72] | 617.79 [501.79 to 760.61] | 264.10 [213.25 to 327.07] | 505.46 [403.79 to 632.74] | 495.42 [398.75 to 615.52] | 624.06 [501.90 to 775.95] | 397.32 [318.64 to 495.42]
  Flu B1 Assay 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 0 | 0 | 0 | 0 | 0 | 0 | 101 | 97 | 121 | 115 | 108 | 116 | 115 | 111
  Flu B1 Assay 1 |  |  |  |  |  |  | 190.37 [149.51 to 242.41] |  |  |  |  |  |  | 277.45 [242.32 to 317.66] | 305.19 [266.47 to 349.53] | 341.88 [302.03 to 386.98] | 487.32 [429.42 to 553.02] | 565.86 [493.20 to 649.22] | 532.34 [465.90 to 608.25] | 546.58 [477.99 to 625.02] | 760.08 [663.75 to 870.39]
  Flu B1 Assay 2: number analyzed (Participants) | 19 | 22 | 22 | 23 | 21 | 24 | 23 | 22 | 19 | 21 | 22 | 18 | 21 | 101 | 97 | 121 | 114 | 108 | 115 | 115 | 111
  Flu B1 Assay 2 | 74.84 [56.27 to 99.55] | 149.88 [115.56 to 194.38] | 154.29 [118.95 to 200.13] | 168.29 [130.47 to 217.08] | 160.05 [122.23 to 209.56] | 150.39 [117.31 to 192.80] | 123.35 [95.54 to 159.25] | 151.48 [116.44 to 197.08] | 133.43 [133.43 to 176.42] | 139.36 [106.62 to 182.14] | 151.53 [116.71 to 196.74] | 161.25 [120.77 to 215.31] | 208.78 [158.86 to 274.40] | 97.37 [80.90 to 117.18] | 114.95 [95.61 to 138.20] | 125.81 [106.21 to 149.04] | 200.28 [168.72 to 237.75] | 173.94 [148.07 to 204.32] | 184.85 [158.02 to 216.23] | 193.96 [165.75 to 226.97] | 258.03 [220.10 to 302.50]
  Flu B2 Assay 1: number analyzed (Participants) | 19 | 22 | 22 | 23 | 21 | 24 | 23 | 22 | 19 | 21 | 22 | 19 | 22 | 101 | 96 | 121 | 115 | 108 | 116 | 115 | 111
  Flu B2 Assay 1 | 240.13 [184.19 to 313.06] | 689.10 [540.89 to 877.93] | 536.73 [421.29 to 683.80] | 727.48 [573.88 to 922.19] | 739.83 [576.07 to 950.14] | 689.88 [547.45 to 869.37] | 536.57 [422.95 to 680.71] | 568.51 [445.35 to 725.73] | 624.12 [481.46 to 809.04] | 617.81 [481.21 to 793.19] | 534.31 [418.77 to 681.73] | 501.11 [386.00 to 650.53] | 764.90 [596.95 to 980.11] | 605.48 [534.15 to 686.34] | 692.40 [610.63 to 785.13] | 687.04 [613.05 to 769.95] | 913.91 [813.27 to 1027.00] | 516.25 [452.96 to 588.38] | 583.05 [513.21 to 662.39] | 621.87 [547.30 to 706.61] | 744.28 [654.26 to 846.70]
  Flu B2 Assay 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 0 | 0 | 0 | 0 | 0 | 0 | 101 | 97 | 121 | 114 | 108 | 115 | 115 | 111
  Flu B2 Assay 2 |  |  |  |  |  |  | 45.65 [31.51 to 66.12] |  |  |  |  |  |  | 370.16 [316.87 to 432.43] | 409.56 [350.40 to 478.70] | 446.20 [387.24 to 514.14] | 440.96 [381.00 to 510.34] | 283.03 [236.19 to 339.15] | 281.44 [235.95 to 335.72] | 299.04 [250.56 to 356.90] | 329.89 [275.95 to 394.36]

10. Primary Outcome: Geometric Mean Increase (GMI) of Antigen 1 Antibody Titers From Day 1 to Day 29
Description: GMI is defined as the geometric mean of the ratios of the post dosing titer over the Day 1 titer. Assay 1= with egg propagated Influenza virus and Assay 2= with cell propagated Influenza virus.
Time Frame: From Day 1 (baseline) to Day 29
Population: The analysis was performed on the PPS. Only participants with data available for the specified analysis at the specified timepoints were included.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Flu mRNA_Ph1_1 Younger Adults (YA) Group | Flu mRNA_Ph1_2 YA Group | Flu mRNA_Ph1_3 YA Group | Flu mRNA_Ph1_4 YA Group | Flu mRNA_Ph1_5 YA Group | Flu mRNA_Ph1_6 YA Group | Flu mRNA_Ph1_7 YA Group | Flu mRNA_Ph1_8 YA Group | Flu mRNA_Ph1_9 YA Group | Flu mRNA_Ph1_10 YA Group | Flu mRNA_Ph1_11 YA Group | Flu mRNA_Ph1_12 YA Group | Control Ph1_YA Group | Flu mRNA_Ph2_1_YA Group | Flu mRNA_Ph2_2_YA Group | Flu mRNA_Ph2_3_YA Group | Control_Ph2_YA Group | Flu mRNA_Ph2_1_Older Adults (OA) Group | Flu mRNA_Ph2_2_OA Group | Flu mRNA_Ph2_3_OA Group | Control_Ph2_OA Group
Number analyzed (Participants) | 19 | 22 | 22 | 23 | 21 | 24 | 23 | 22 | 19 | 21 | 22 | 19 | 22 | 101 | 97 | 121 | 115 | 108 | 116 | 115 | 111
Ratio
  Flu A1 Assay 1: number analyzed (Participants) | 19 | 22 | 22 | 23 | 21 | 24 | 23 | 22 | 19 | 21 | 22 | 19 | 22 | 101 | 92 | 119 | 114 | 107 | 112 | 113 | 111
  Flu A1 Assay 1 | 12.83 [8.21 to 20.04] | 9.16 [6.09 to 13.77] | 6.77 [4.50 to 10.18] | 9.81 [6.58 to 14.63] | 10.39 [6.82 to 15.84] | 9.06 [6.13 to 13.40] | 9.54 [6.38 to 14.26] | 8.86 [5.87 to 13.36] | 11.20 [7.24 to 17.33] | 10.12 [6.65 to 15.39] | 8.42 [5.58 to 12.70] | 9.32 [6.01 to 14.46] | 6.14 [4.05 to 9.31] | 6.42 [5.06 to 8.16] | 7.89 [6.19 to 10.06] | 9.51 [7.63 to 11.84] | 5.92 [4.73 to 7.40] | 6.34 [4.97 to 8.09] | 8.59 [6.77 to 10.90] | 9.53 [7.51 to 12.10] | 5.99 [4.72 to 7.60]
  Flu A1 Assay 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 0 | 0 | 0 | 0 | 0 | 0 | 101 | 97 | 121 | 114 | 108 | 115 | 115 | 111
  Flu A1 Assay 2 |  |  |  |  |  |  | 6.33 [3.96 to 10.12] |  |  |  |  |  |  | 5.36 [4.26 to 6.74] | 5.32 [4.23 to 6.69] | 5.96 [4.84 to 7.35] | 3.58 [2.89 to 4.44] | 4.20 [3.32 to 5.30] | 4.72 [3.76 to 5.92] | 5.56 [4.42 to 6.99] | 2.90 [2.30 to 3.65]
  Flu A2 Assay 1 | 1.32 [0.84 to 2.05] | 11.41 [7.60 to 17.11] | 7.61 [5.07 to 11.41] | 12.08 [8.12 to 17.96] | 7.39 [4.86 to 11.24] | 8.26 [5.60 to 12.19] | 7.38 [4.96 to 11.00] | 8.21 [5.45 to 12.36] | 9.26 [5.99 to 14.32] | 8.39 [5.52 to 12.74] | 11.38 [7.58 to 17.11] | 7.44 [4.81 to 11.53] | 3.20 [2.11 to 4.84] | 6.92 [5.57 to 8.60] | 7.96 [6.41 to 9.90] | 10.09 [8.27 to 12.30] | 4.13 [3.37 to 5.06] | 8.35 [6.68 to 10.43] | 8.41 [6.78 to 10.44] | 10.00 [8.05 to 12.43] | 5.62 [4.51 to 7.00]
  Flu A2 Assay 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 0 | 19 | 0 | 0 | 0 | 0 | 101 | 97 | 121 | 114 | 108 | 115 | 115 | 111
  Flu A2 Assay 2 |  |  |  |  |  |  | 4.62 [2.85 to 7.48] |  | 14.87 [8.87 to 24.93] |  |  |  |  | 3.75 [2.99 to 4.71] | 4.04 [3.21 to 5.08] | 5.32 [4.32 to 6.55] | 2.27 [1.84 to 2.82] | 3.24 [2.59 to 4.06] | 3.18 [2.56 to 3.95] | 4.00 [3.22 to 4.98] | 2.55 [2.04 to 3.18]
  Flu B1 Assay 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 0 | 0 | 0 | 0 | 0 | 0 | 101 | 97 | 121 | 115 | 108 | 116 | 115 | 111
  Flu B1 Assay 1 |  |  |  |  |  |  | 1.64 [1.29 to 2.09] |  |  |  |  |  |  | 1.40 [1.22 to 1.60] | 1.54 [1.35 to 1.77] | 1.73 [1.53 to 1.95] | 2.46 [2.17 to 2.79] | 2.51 [2.19 to 2.88] | 2.36 [2.07 to 2.70] | 2.43 [2.12 to 2.77] | 3.37 [2.94 to 3.86]
  Flu B1 Assay 2: number analyzed (Participants) | 19 | 22 | 22 | 23 | 21 | 24 | 23 | 22 | 19 | 21 | 22 | 18 | 21 | 101 | 97 | 121 | 114 | 108 | 115 | 115 | 111
  Flu B1 Assay 2 | 0.93 [0.70 to 1.24] | 1.87 [1.44 to 2.42] | 1.92 [1.48 to 2.49] | 2.09 [1.62 to 2.70] | 1.99 [1.52 to 2.61] | 1.87 [1.46 to 2.40] | 1.54 [1.19 to 1.98] | 1.89 [1.45 to 2.45] | 1.66 [1.26 to 2.20] | 1.73 [1.33 to 2.27] | 1.89 [1.45 to 2.45] | 2.01 [1.50 to 2.68] | 2.60 [1.98 to 3.41] | 1.83 [1.52 to 2.20] | 2.16 [1.80 to 2.60] | 2.36 [2.00 to 2.80] | 3.76 [3.17 to 4.47] | 1.77 [1.51 to 2.08] | 1.89 [1.61 to 2.21] | 1.98 [1.69 to 2.32] | 2.63 [2.25 to 3.09]
  Flu B2 Assay 1: number analyzed (Participants) | 19 | 22 | 22 | 23 | 21 | 24 | 23 | 22 | 19 | 21 | 22 | 19 | 22 | 101 | 96 | 121 | 115 | 108 | 116 | 115 | 111
  Flu B2 Assay 1 | 1.09 [0.84 to 1.42] | 3.13 [2.45 to 3.98] | 2.43 [1.91 to 3.10] | 3.30 [2.60 to 4.18] | 3.36 [2.61 to 4.31] | 3.13 [2.48 to 3.94] | 2.43 [1.92 to 3.09] | 2.58 [2.02 to 3.29] | 2.83 [2.18 to 3.67] | 2.80 [2.18 to 3.60] | 2.42 [1.90 to 3.09] | 2.27 [1.75 to 2.95] | 3.47 [2.71 to 4.45] | 2.04 [1.80 to 2.31] | 2.33 [2.06 to 2.64] | 2.31 [2.06 to 2.59] | 3.08 [2.74 to 3.46] | 2.40 [2.10 to 2.73] | 2.71 [2.38 to 3.08] | 2.89 [2.54 to 3.28] | 3.46 [3.04 to 3.93]
  Flu B2 Assay 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 0 | 0 | 0 | 0 | 0 | 0 | 101 | 97 | 121 | 114 | 108 | 115 | 115 | 111
  Flu B2 Assay 2 |  |  |  |  |  |  | 3.18 [2.20 to 4.61] |  |  |  |  |  |  | 1.72 [1.47 to 2.01] | 1.90 [1.63 to 2.22] | 2.07 [1.80 to 2.39] | 2.05 [1.77 to 2.37] | 1.39 [1.16 to 1.66] | 1.38 [1.16 to 1.65] | 1.47 [1.23 to 1.75] | 1.62 [1.35 to 1.94]

11. Primary Outcome: Percentage of Participants With Antigen 1 Antibody Seroconversion Rate (SCR)
Description: SCR is defined as the percentage of dosed participants who have either an anti-vaccine antibody pre-dose titer < 1:10 and a post-dose anti-vaccine antibody titer >= 1:40 or a pre-dose anti-vaccine antibody titer >= 1:10 and at least a 4-fold increase in post-dose anti-vaccine antibody titer. Assay 1= with egg propagated Influenza virus and Assay 2= with cell propagated Influenza virus.
Time Frame: From Day 1 to Day 29
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Flu mRNA_Ph1_1 Younger Adults (YA) Group | Flu mRNA_Ph1_2 YA Group | Flu mRNA_Ph1_3 YA Group | Flu mRNA_Ph1_4 YA Group | Flu mRNA_Ph1_5 YA Group | Flu mRNA_Ph1_6 YA Group | Flu mRNA_Ph1_7 YA Group | Flu mRNA_Ph1_8 YA Group | Flu mRNA_Ph1_9 YA Group | Flu mRNA_Ph1_10 YA Group | Flu mRNA_Ph1_11 YA Group | Flu mRNA_Ph1_12 YA Group | Control Ph1_YA Group | Flu mRNA_Ph2_1_YA Group | Flu mRNA_Ph2_2_YA Group | Flu mRNA_Ph2_3_YA Group | Control_Ph2_YA Group | Flu mRNA_Ph2_1_Older Adults (OA) Group | Flu mRNA_Ph2_2_OA Group | Flu mRNA_Ph2_3_OA Group | Control_Ph2_OA Group
Number analyzed (Participants) | 19 | 22 | 22 | 23 | 21 | 24 | 23 | 22 | 19 | 21 | 22 | 19 | 22 | 101 | 97 | 121 | 115 | 108 | 116 | 115 | 111
Percentage of participants
  Flu A1 Assay 1: number analyzed (Participants) | 19 | 22 | 22 | 23 | 21 | 24 | 23 | 22 | 19 | 21 | 22 | 19 | 22 | 101 | 94 | 119 | 114 | 107 | 112 | 113 | 111
  Flu A1 Assay 1 | 78.9 [54.4 to 93.9] | 68.2 [45.1 to 86.1] | 59.1 [36.4 to 79.3] | 65.2 [42.7 to 83.6] | 57.1 [34.0 to 78.2] | 70.8 [48.9 to 87.4] | 60.9 [38.5 to 80.3] | 63.6 [40.7 to 82.8] | 73.7 [48.8 to 90.9] | 81.0 [58.1 to 94.6] | 68.2 [45.1 to 86.1] | 57.9 [33.5 to 79.7] | 59.1 [36.4 to 79.3] | 49.5 [39.4 to 59.6] | 63.8 [53.3 to 73.5] | 67.2 [58.0 to 75.6] | 47.4 [37.9 to 56.9] | 51.4 [41.5 to 61.2] | 63.4 [53.8 to 72.3] | 64.6 [55.0 to 73.4] | 49.5 [39.9 to 59.2]
  Flu A1 Assay 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 0 | 0 | 0 | 0 | 0 | 0 | 101 | 97 | 121 | 114 | 108 | 115 | 115 | 111
  Flu A1 Assay 2 |  |  |  |  |  |  | 56.5 [34.5 to 76.8] |  |  |  |  |  |  | 60.4 [50.2 to 70.0] | 62.9 [52.5 to 72.5] | 62.8 [53.6 to 71.4] | 50.0 [40.5 to 59.5] | 49.1 [39.3 to 58.9] | 59.1 [49.6 to 68.2] | 60.9 [51.3 to 69.8] | 36.0 [27.1 to 45.7]
  Flu A2 Assay 1 | 5.3 [0.1 to 26.0] | 90.9 [70.8 to 98.9] | 68.2 [45.1 to 86.1] | 87.0 [66.4 to 97.2] | 71.4 [47.8 to 88.7] | 79.2 [57.8 to 92.9] | 73.9 [51.6 to 89.8] | 68.2 [45.1 to 86.1] | 68.4 [43.4 to 87.4] | 90.5 [69.6 to 98.8] | 77.3 [54.6 to 92.2] | 47.4 [24.4 to 71.1] | 31.8 [13.9 to 54.9] | 72.3 [62.5 to 80.7] | 70.1 [60.0 to 79.0] | 79.3 [71.0 to 86.2] | 38.3 [29.4 to 47.8] | 62.0 [52.2 to 71.2] | 69.0 [59.7 to 77.2] | 71.3 [62.1 to 79.4] | 54.1 [44.3 to 63.6]
  Flu A2 Assay 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 0 | 19 | 0 | 0 | 0 | 0 | 101 | 97 | 121 | 114 | 108 | 115 | 115 | 111
  Flu A2 Assay 2 |  |  |  |  |  |  | 65.2 [42.7 to 83.6] |  | 84.2 [60.4 to 96.6] |  |  |  |  | 54.5 [44.2 to 64.4] | 49.5 [39.2 to 59.8] | 63.6 [54.4 to 72.2] | 37.7 [28.8 to 47.3] | 43.5 [34.0 to 53.4] | 52.2 [42.7 to 61.6] | 53.9 [44.4 to 63.2] | 38.7 [29.6 to 48.5]
  Flu B1 Assay 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 0 | 0 | 0 | 0 | 0 | 0 | 101 | 97 | 121 | 115 | 108 | 116 | 115 | 111
  Flu B1 Assay 1 |  |  |  |  |  |  | 8.7 [1.1 to 28.0] |  |  |  |  |  |  | 12.9 [7.0 to 21.0] | 12.4 [6.6 to 20.6] | 17.4 [11.1 to 25.3] | 32.2 [23.8 to 41.5] | 28.7 [20.4 to 38.2] | 27.6 [19.7 to 36.7] | 29.6 [21.4 to 38.8] | 41.4 [32.2 to 51.2]
  Flu B1 Assay 2: number analyzed (Participants) | 19 | 22 | 22 | 23 | 21 | 24 | 23 | 22 | 19 | 21 | 22 | 18 | 21 | 101 | 97 | 121 | 114 | 108 | 115 | 115 | 111
  Flu B1 Assay 2 | 0 [0 to 17.6] | 13.6 [2.9 to 34.9] | 22.7 [7.8 to 45.4] | 17.4 [5.0 to 38.8] | 19.0 [5.4 to 41.9] | 16.7 [4.7 to 37.4] | 4.3 [0.1 to 21.9] | 13.6 [2.9 to 34.9] | 10.5 [1.3 to 33.1] | 19.0 [5.4 to 41.9] | 18.2 [5.2 to 40.3] | 16.7 [3.6 to 41.4] | 33.3 [14.6 to 57.0] | 12.9 [7.0 to 21.0] | 20.6 [13.1 to 30.0] | 19.0 [12.4 to 27.1] | 43.9 [34.6 to 53.5] | 17.6 [10.9 to 26.1] | 22.6 [15.3 to 31.3] | 20.9 [13.9 to 29.4] | 32.4 [23.9 to 42.0]
  Flu B2 Assay 1: number analyzed (Participants) | 19 | 22 | 22 | 23 | 21 | 24 | 23 | 22 | 19 | 21 | 22 | 19 | 22 | 101 | 96 | 121 | 115 | 108 | 116 | 115 | 111
  Flu B2 Assay 1 | 0 [0 to 17.6] | 36.4 [17.2 to 59.3] | 27.3 [10.7 to 50.2] | 52.2 [30.6 to 73.2] | 47.6 [25.7 to 70.2] | 33.3 [15.6 to 55.3] | 26.1 [10.2 to 48.4] | 18.2 [5.2 to 40.3] | 31.6 [12.6 to 56.6] | 47.6 [25.7 to 70.2] | 27.3 [10.7 to 50.2] | 15.8 [3.4 to 39.6] | 54.5 [32.2 to 75.6] | 25.7 [17.6 to 35.4] | 26.0 [17.6 to 36.0] | 23.1 [16.0 to 31.7] | 36.5 [27.7 to 46.0] | 38.0 [28.8 to 47.8] | 38.8 [29.9 to 48.3] | 40.9 [31.8 to 50.4] | 39.6 [30.5 to 49.4]
  Flu B2 Assay 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 0 | 0 | 0 | 0 | 0 | 0 | 101 | 97 | 121 | 114 | 108 | 115 | 115 | 111
  Flu B2 Assay 2 |  |  |  |  |  |  | 26.1 [10.2 to 48.4] |  |  |  |  |  |  | 17.8 [10.9 to 26.7] | 21.6 [13.9 to 31.2] | 24.0 [16.7 to 32.6] | 21.9 [14.7 to 30.6] | 17.6 [10.9 to 26.1] | 20.0 [13.1 to 28.5] | 17.4 [11.0 to 25.6] | 23.4 [15.9 to 32.4]

12. Primary Outcome: Percentage of Participants With Antigen 1 Antibody Seroprotection Rate (SPR)
Description: SPR is defined as the percentage of dosed participants with a anti-vaccine antibody titer >= 1:40. Assay 1= with egg propagated Influenza virus and Assay 2= with cell propagated Influenza virus.
Time Frame: At Day 1
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Flu mRNA_Ph1_1 Younger Adults (YA) Group | Flu mRNA_Ph1_2 YA Group | Flu mRNA_Ph1_3 YA Group | Flu mRNA_Ph1_4 YA Group | Flu mRNA_Ph1_5 YA Group | Flu mRNA_Ph1_6 YA Group | Flu mRNA_Ph1_7 YA Group | Flu mRNA_Ph1_8 YA Group | Flu mRNA_Ph1_9 YA Group | Flu mRNA_Ph1_10 YA Group | Flu mRNA_Ph1_11 YA Group | Flu mRNA_Ph1_12 YA Group | Control Ph1_YA Group | Flu mRNA_Ph2_1_YA Group | Flu mRNA_Ph2_2_YA Group | Flu mRNA_Ph2_3_YA Group | Control_Ph2_YA Group | Flu mRNA_Ph2_1_Older Adults (OA) Group | Flu mRNA_Ph2_2_OA Group | Flu mRNA_Ph2_3_OA Group | Control_Ph2_OA Group
Number analyzed (Participants) | 20 | 22 | 22 | 23 | 21 | 24 | 23 | 22 | 21 | 21 | 22 | 21 | 22 | 102 | 99 | 125 | 116 | 110 | 117 | 119 | 117
Percentage of participants
  Flu A1 Assay 1: number analyzed (Participants) | 20 | 22 | 22 | 23 | 21 | 24 | 23 | 22 | 21 | 21 | 22 | 21 | 22 | 102 | 96 | 123 | 115 | 110 | 114 | 116 | 117
  Flu A1 Assay 1 | 60.0 [36.1 to 80.9] | 63.6 [40.7 to 82.8] | 50.0 [28.2 to 71.8] | 65.2 [42.7 to 83.6] | 61.9 [38.4 to 81.9] | 37.5 [18.8 to 59.4] | 69.6 [47.1 to 86.8] | 54.5 [32.2 to 75.6] | 66.7 [43.0 to 85.4] | 47.6 [25.7 to 70.2] | 45.5 [24.4 to 67.8] | 47.6 [25.7 to 70.2] | 45.5 [24.4 to 67.8] | 13.7 [7.7 to 22.0] | 8.3 [3.7 to 15.8] | 7.3 [3.4 to 13.4] | 9.6 [4.9 to 16.5] | 13.6 [7.8 to 21.5] | 14.9 [8.9 to 22.8] | 8.6 [4.2 to 15.3] | 16.2 [10.1 to 24.2]
  Flu A1 Assay 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 0 | 0 | 0 | 0 | 0 | 0 | 102 | 99 | 125 | 116 | 110 | 117 | 119 | 117
  Flu A1 Assay 2 |  |  |  |  |  |  | 34.8 [16.4 to 57.3] |  |  |  |  |  |  | 70.6 [60.7 to 79.2] | 71.7 [61.8 to 80.3] | 66.4 [57.4 to 74.6] | 60.3 [50.8 to 69.3] | 84.5 [76.4 to 90.7] | 71.8 [62.7 to 79.7] | 65.5 [56.3 to 74.0] | 88.9 [81.7 to 93.9]
  Flu A2 Assay 1 | 20.0 [5.7 to 43.7] | 27.3 [10.7 to 50.2] | 22.7 [7.8 to 45.4] | 13.0 [2.8 to 33.6] | 33.3 [14.6 to 57.0] | 8.3 [1.0 to 27.0] | 26.1 [10.2 to 48.4] | 36.4 [17.2 to 59.3] | 33.3 [14.6 to 57.0] | 9.5 [1.2 to 30.4] | 27.3 [10.7 to 50.2] | 28.6 [11.3 to 52.2] | 27.3 [10.7 to 50.2] | 18.6 [11.6 to 27.6] | 22.2 [14.5 to 31.7] | 21.6 [14.7 to 29.8] | 32.8 [24.3 to 42.1] | 38.2 [29.1 to 47.9] | 30.8 [22.6 to 40.0] | 31.9 [23.7 to 41.1] | 32.5 [24.1 to 41.8]
  Flu A2 Assay 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 0 | 21 | 0 | 0 | 0 | 0 | 102 | 99 | 125 | 116 | 110 | 117 | 119 | 117
  Flu A2 Assay 2 |  |  |  |  |  |  | 78.3 [56.3 to 92.5] |  | 81.0 [58.1 to 94.6] |  |  |  |  | 78.4 [69.2 to 86.0] | 78.8 [69.4 to 86.4] | 77.6 [69.3 to 84.6] | 82.8 [74.6 to 89.1] | 91.8 [85.0 to 96.2] | 86.3 [78.7 to 92.0] | 82.4 [74.3 to 88.7] | 88.9 [81.7 to 93.9]
  Flu B1 Assay 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 0 | 0 | 0 | 0 | 0 | 0 | 102 | 99 | 125 | 116 | 110 | 117 | 119 | 117
  Flu B1 Assay 1 |  |  |  |  |  |  | 100 [85.2 to 100] |  |  |  |  |  |  | 97.1 [91.6 to 99.4] | 98.0 [92.9 to 99.8] | 98.4 [94.3 to 99.8] | 96.6 [91.4 to 99.1] | 93.6 [87.3 to 97.4] | 94.9 [89.2 to 98.1] | 99.2 [95.4 to 100] | 99.1 [95.3 to 100]
  Flu B1 Assay 2: number analyzed (Participants) | 20 | 22 | 22 | 23 | 21 | 24 | 23 | 22 | 21 | 21 | 22 | 20 | 21 | 102 | 99 | 125 | 116 | 110 | 117 | 119 | 117
  Flu B1 Assay 2 | 85.0 [62.1 to 96.8] | 95.5 [77.2 to 99.9] | 86.4 [65.1 to 97.1] | 95.7 [78.1 to 99.9] | 76.2 [52.8 to 91.8] | 91.7 [73.0 to 99.0] | 95.7 [78.1 to 99.9] | 95.5 [77.2 to 99.9] | 100 [83.9 to 100] | 76.2 [52.8 to 91.8] | 100 [84.6 to 100] | 95.0 [75.1 to 99.9] | 85.7 [63.7 to 97.0] | 71.6 [61.8 to 80.1] | 68.7 [58.6 to 77.6] | 62.4 [53.3 to 70.9] | 63.8 [54.4 to 72.5] | 83.6 [75.4 to 90.0] | 81.2 [72.9 to 87.8] | 84.9 [77.2 to 90.8] | 86.3 [78.7 to 92.0]
  Flu B2 Assay 1: number analyzed (Participants) | 20 | 22 | 22 | 23 | 21 | 24 | 23 | 22 | 21 | 21 | 22 | 21 | 22 | 102 | 98 | 125 | 116 | 110 | 117 | 119 | 117
  Flu B2 Assay 1 | 100 [83.2 to 100] | 95.5 [77.2 to 99.9] | 100 [84.6 to 100] | 100 [85.2 to 100] | 100 [83.9 to 100] | 100 [85.8 to 100] | 100 [85.2 to 100] | 100 [84.6 to 100] | 100 [83.9 to 100] | 100 [83.9 to 100] | 100 [84.6 to 100] | 95.2 [76.2 to 99.9] | 95.5 [77.2 to 99.9] | 97.1 [91.6 to 99.4] | 100 [96.3 to 100] | 100 [97.1 to 100] | 99.1 [95.3 to 100] | 95.5 [89.7 to 98.5] | 98.3 [94.0 to 99.8] | 97.5 [92.8 to 99.5] | 99.1 [95.3 to 100]
  Flu B2 Assay 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 0 | 0 | 0 | 0 | 0 | 0 | 102 | 99 | 125 | 116 | 110 | 117 | 119 | 117
  Flu B2 Assay 2 |  |  |  |  |  |  | 26.1 [10.2 to 48.4] |  |  |  |  |  |  | 98.0 [93.1 to 99.8] | 96.0 [90.0 to 98.9] | 97.6 [93.1 to 99.5] | 98.3 [93.9 to 99.8] | 96.4 [91.0 to 99.0] | 95.7 [90.3 to 98.6] | 95.0 [89.3 to 98.1] | 98.3 [94.0 to 99.8]

13. Primary Outcome: Percentage of Participants With Antigen 1 Antibody SPR
Description: Assay 1= with egg propagated Influenza virus and Assay 2= with cell propagated Influenza virus.
Time Frame: At Day 29
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Flu mRNA_Ph1_1 Younger Adults (YA) Group | Flu mRNA_Ph1_2 YA Group | Flu mRNA_Ph1_3 YA Group | Flu mRNA_Ph1_4 YA Group | Flu mRNA_Ph1_5 YA Group | Flu mRNA_Ph1_6 YA Group | Flu mRNA_Ph1_7 YA Group | Flu mRNA_Ph1_8 YA Group | Flu mRNA_Ph1_9 YA Group | Flu mRNA_Ph1_10 YA Group | Flu mRNA_Ph1_11 YA Group | Flu mRNA_Ph1_12 YA Group | Control Ph1_YA Group | Flu mRNA_Ph2_1_YA Group | Flu mRNA_Ph2_2_YA Group | Flu mRNA_Ph2_3_YA Group | Control_Ph2_YA Group | Flu mRNA_Ph2_1_Older Adults (OA) Group | Flu mRNA_Ph2_2_OA Group | Flu mRNA_Ph2_3_OA Group | Control_Ph2_OA Group
Number analyzed (Participants) | 19 | 22 | 22 | 23 | 21 | 24 | 23 | 22 | 19 | 21 | 22 | 19 | 22 | 101 | 97 | 121 | 115 | 108 | 116 | 115 | 111
Percentage of participants
  Flu A1 Assay 1: number analyzed (Participants) | 19 | 22 | 22 | 23 | 21 | 24 | 23 | 22 | 19 | 21 | 22 | 19 | 22 | 101 | 96 | 120 | 115 | 107 | 112 | 115 | 111
  Flu A1 Assay 1 | 94.7 [74.0 to 99.9] | 100 [84.6 to 100] | 90.9 [70.8 to 98.9] | 100 [85.2 to 100] | 100 [83.9 to 100] | 95.8 [78.9 to 99.9] | 95.7 [78.1 to 99.9] | 95.5 [77.2 to 99.9] | 94.7 [74.0 to 99.9] | 95.2 [76.2 to 99.9] | 95.5 [77.2 to 99.9] | 100 [82.4 to 100] | 95.5 [77.2 to 99.9] | 55.4 [45.2 to 65.3] | 65.6 [55.2 to 75.0] | 73.3 [64.5 to 81.0] | 63.5 [54.0 to 72.3] | 64.5 [54.6 to 73.5] | 72.3 [63.1 to 80.4] | 71.3 [62.1 to 79.4] | 69.4 [59.9 to 77.8]
  Flu A1 Assay 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 0 | 0 | 0 | 0 | 0 | 0 | 101 | 97 | 121 | 114 | 108 | 115 | 115 | 111
  Flu A1 Assay 2 |  |  |  |  |  |  | 82.6 [61.2 to 95.0] |  |  |  |  |  |  | 95.0 [88.8 to 98.4] | 95.9 [89.8 to 98.9] | 99.2 [95.5 to 100] | 87.7 [80.3 to 93.1] | 97.2 [92.1 to 99.4] | 94.8 [89.0 to 98.1] | 96.5 [91.3 to 99.0] | 90.1 [83.0 to 94.9]
  Flu A2 Assay 1 | 31.6 [12.6 to 56.6] | 100 [84.6 to 100] | 72.7 [49.8 to 89.3] | 95.7 [78.1 to 99.9] | 90.5 [69.6 to 98.8] | 79.2 [57.8 to 92.9] | 82.6 [61.2 to 95.0] | 90.9 [70.8 to 98.9] | 89.5 [66.9 to 98.7] | 95.2 [76.2 to 99.9] | 86.4 [65.1 to 97.1] | 84.2 [60.4 to 96.6] | 59.1 [36.4 to 79.3] | 83.2 [74.4 to 89.9] | 83.5 [74.6 to 90.3] | 92.6 [86.3 to 96.5] | 69.6 [60.3 to 77.8] | 88.0 [80.3 to 93.4] | 86.2 [78.6 to 91.9] | 90.4 [83.5 to 95.1] | 81.1 [72.5 to 87.9]
  Flu A2 Assay 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 0 | 19 | 0 | 0 | 0 | 0 | 101 | 97 | 121 | 114 | 108 | 115 | 115 | 111
  Flu A2 Assay 2 |  |  |  |  |  |  | 100 [85.2 to 100] |  | 100 [82.4 to 100] |  |  |  |  | 100 [96.4 to 100] | 99.0 [94.4 to 100] | 100 [97.0 to 100] | 98.2 [93.8 to 99.8] | 100 [96.6 to 100] | 98.3 [93.9 to 99.8] | 100 [96.8 to 100] | 97.3 [92.3 to 99.4]
  Flu B1 Assay 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 0 | 0 | 0 | 0 | 0 | 0 | 101 | 97 | 121 | 115 | 108 | 116 | 115 | 111
  Flu B1 Assay 1 |  |  |  |  |  |  | 100 [85.2 to 100] |  |  |  |  |  |  | 99.0 [94.6 to 100] | 97.9 [92.7 to 99.7] | 99.2 [95.5 to 100] | 100 [96.8 to 100] | 100 [96.6 to 100] | 100 [96.9 to 100] | 99.1 [95.3 to 100] | 100 [96.7 to 100]
  Flu B1 Assay 2: number analyzed (Participants) | 19 | 22 | 22 | 23 | 21 | 24 | 23 | 22 | 19 | 21 | 22 | 19 | 22 | 101 | 97 | 121 | 114 | 108 | 115 | 115 | 111
  Flu B1 Assay 2 | 84.2 [60.4 to 96.6] | 100 [86.6 to 100] | 95.4 [77.2 to 99.9] | 100 [85.2 to 100] | 100 [83.9 to 100] | 100 [85.8 to 100] | 100 [85.2 to 100] | 100 [84.6 to 100] | 100 [82.4 to 100] | 95.2 [76.2 to 99.9] | 100 [84.6 to 100] | 100 [82.4 to 100] | 100 [84.6 to 100] | 82.2 [73.3 to 89.1] | 83.5 [74.6 to 90.3] | 83.5 [75.6 to 89.6] | 95.6 [90.1 to 98.6] | 97.2 [92.1 to 99.4] | 96.5 [91.3 to 99.0] | 97.4 [92.6 to 99.5] | 100 [96.7 to 100]
  Flu B2 Assay 1: number analyzed (Participants) | 19 | 22 | 22 | 23 | 21 | 24 | 23 | 22 | 19 | 21 | 22 | 19 | 22 | 101 | 96 | 121 | 115 | 108 | 116 | 115 | 111
  Flu B2 Assay 1 | 100 [82.4 to 100] | 100 [84.6 to 100] | 100 [84.6 to 100] | 100 [85.2 to 100] | 100 [83.9 to 100] | 100 [85.8 to 100] | 100 [85.2 to 100] | 100 [84.6 to 100] | 100 [82.4 to 100] | 100 [83.9 to 100] | 100 [84.6 to 100] | 100 [82.4 to 100] | 100 [84.6 to 100] | 100 [96.4 to 100] | 100 [96.2 to 100] | 100 [97.0 to 100] | 100 [96.8 to 100] | 100 [96.6 to 100] | 100 [96.9 to 100] | 100 [96.8 to 100] | 100 [96.7 to 100]
  Flu B2 Assay 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 0 | 0 | 0 | 0 | 0 | 0 | 101 | 97 | 121 | 114 | 108 | 115 | 115 | 111
  Flu B2 Assay 2 |  |  |  |  |  |  | 56.5 [34.5 to 76.8] |  |  |  |  |  |  | 100 [96.4 to 100] | 99.0 [94.4 to 100] | 100 [97.0 to 100] | 100 [96.8 to 100] | 98.1 [93.5 to 99.8] | 99.1 [95.3 to 100] | 99.1 [95.3 to 100] | 98.2 [93.6 to 99.8]

14. Primary Outcome: GMT of Antigen 2 Antibody Titer
Time Frame: At Day 29
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Flu mRNA_Ph1_1 Younger Adults (YA) Group | Flu mRNA_Ph1_2 YA Group | Flu mRNA_Ph1_3 YA Group | Flu mRNA_Ph1_4 YA Group | Flu mRNA_Ph1_5 YA Group | Flu mRNA_Ph1_6 YA Group | Flu mRNA_Ph1_7 YA Group | Flu mRNA_Ph1_8 YA Group | Flu mRNA_Ph1_9 YA Group | Flu mRNA_Ph1_10 YA Group | Flu mRNA_Ph1_11 YA Group | Flu mRNA_Ph1_12 YA Group | Control Ph1_YA Group | Flu mRNA_Ph2_1_YA Group | Flu mRNA_Ph2_2_YA Group | Flu mRNA_Ph2_3_YA Group | Control_Ph2_YA Group | Flu mRNA_Ph2_1_Older Adults (OA) Group | Flu mRNA_Ph2_2_OA Group | Flu mRNA_Ph2_3_OA Group | Control_Ph2_OA Group
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 22 | 19 | 21 | 22 | 19 | 22 | 101 | 97 | 121 | 115 | 108 | 116 | 115 | 111
Titers
  Flu A1 |  |  |  |  |  |  | 5588.80 [4242.15 to 7362.94] | 4087.84 [3073.11 to 5437.63] | 4140.51 [3070.75 to 5582.93] | 5830.63 [4362.90 to 7792.13] | 5311.18 [4005.78 to 7041.98] | 6374.69 [4720.97 to 8607.68] | 1126.63 [840.59 to 1510.00] | 763.90 [652.50 to 894.32] | 940.60 [802.48 to 1102.49] | 988.40 [855.52 to 1141.91] | 151.87 [131.07 to 175.97] | 863.96 [733.17 to 1018.07] | 835.61 [712.72 to 979.69] | 1159.00 [987.31 to 1360.55] | 194.60 [165.47 to 228.85]
  Flu A2 |  |  |  |  |  |  | 782.28 [634.47 to 964.53] | 974.11 [783.89 to 1210.50] | 755.19 [602.64 to 946.35] | 868.89 [694.91 to 1086.43] | 984.15 [794.34 to 1219.31] | 1137.13 [902.89 to 1432.13] | 424.76 [339.51 to 531.43] | 778.89 [686.52 to 883.69] | 920.46 [810.96 to 1044.75] | 1070.07 [952.77 to 1201.82] | 369.35 [328.29 to 415.54] | 1107.49 [967.90 to 1267.21] | 1156.39 [1014.68 to 1317.91] | 1355.41 [1188.24 to 1546.10] | 504.28 [441.44 to 576.06]
  Flu B1 |  |  |  |  |  |  | 1494.07 [1135.89 to 1965.20] | 2122.26 [1599.71 to 2815.50] | 1693.64 [1259.15 to 2278.06] | 1673.20 [1256.77 to 2227.62] | 1459.78 [1103.36 to 1931.34] | 1903.93 [1409.82 to 2571.23] | 926.76 [692.23 to 1240.76] | 591.78 [519.62 to 673.97] | 696.93 [612.01 to 793.65] | 763.06 [677.81 to 859.03] | 376.75 [333.71 to 425.33] | 719.59 [624.28 to 829.45] | 759.26 [661.67 to 871.25] | 941.93 [819.50 to 1082.65] | 483.95 [420.71 to 556.70]
  Flu B2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 22 | 19 | 21 | 22 | 18 | 22 | 101 | 96 | 120 | 115 | 108 | 116 | 115 | 111
  Flu B2 |  |  |  |  |  |  | 2566.54 [1990.57 to 3309.17] | 3373.58 [2593.73 to 4387.90] | 3214.91 [2441.12 to 4233.98] | 3281.89 [2515.38 to 4281.98] | 2614.82 [2016.67 to 3390.38] | 3204.51 [2412.86 to 4255.89] | 1424.37 [1086.67 to 1867.01] | 2600.03 [2325.91 to 2906.44] | 2911.06 [2600.25 to 3259.02] | 3171.75 [2863.73 to 3512.90] | 1267.32 [1141.86 to 1406.56] | 3405.35 [3042.32 to 3811.71] | 3653.30 [3274.24 to 4076.25] | 4243.16 [3798.55 to 4739.81] | 1999.75 [1788.70 to 2235.72]

15. Primary Outcome: GMI of Antigen 2 Antibody Titer From Day 1 to Day 29
Time Frame: From Day 1 (baseline) to Day 29
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Flu mRNA_Ph1_1 Younger Adults (YA) Group | Flu mRNA_Ph1_2 YA Group | Flu mRNA_Ph1_3 YA Group | Flu mRNA_Ph1_4 YA Group | Flu mRNA_Ph1_5 YA Group | Flu mRNA_Ph1_6 YA Group | Flu mRNA_Ph1_7 YA Group | Flu mRNA_Ph1_8 YA Group | Flu mRNA_Ph1_9 YA Group | Flu mRNA_Ph1_10 YA Group | Flu mRNA_Ph1_11 YA Group | Flu mRNA_Ph1_12 YA Group | Control Ph1_YA Group | Flu mRNA_Ph2_1_YA Group | Flu mRNA_Ph2_2_YA Group | Flu mRNA_Ph2_3_YA Group | Control_Ph2_YA Group | Flu mRNA_Ph2_1_Older Adults (OA) Group | Flu mRNA_Ph2_2_OA Group | Flu mRNA_Ph2_3_OA Group | Control_Ph2_OA Group
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 22 | 19 | 21 | 22 | 19 | 22 | 101 | 97 | 121 | 115 | 108 | 116 | 115 | 111
Ratio
  Flu A1 |  |  |  |  |  |  | 6.99 [5.31 to 9.22] | 5.12 [3.85 to 6.81] | 5.18 [3.84 to 6.99] | 7.30 [5.46 to 9.75] | 6.65 [5.01 to 8.81] | 7.98 [5.91 to 10.77] | 1.41 [1.05 to 1.89] | 6.37 [5.44 to 7.45] | 7.84 [6.69 to 9.19] | 8.24 [7.13 to 9.52] | 1.27 [1.09 to 1.47] | 6.06 [5.14 to 7.14] | 5.86 [5.00 to 6.87] | 8.13 [6.92 to 9.54] | 1.36 [1.16 to 1.60]
  Flu A2 |  |  |  |  |  |  | 4.00 [3.24 to 4.93] | 4.98 [4.01 to 6.19] | 3.86 [3.08 to 4.84] | 4.44 [3.55 to 5.56] | 5.03 [4.06 to 6.24] | 5.82 [4.62 to 7.32] | 2.17 [1.74 to 2.72] | 3.25 [2.87 to 3.69] | 3.84 [3.39 to 4.36] | 4.47 [3.98 to 5.02] | 1.54 [1.37 to 1.74] | 3.34 [2.92 to 3.82] | 3.49 [3.06 to 3.98] | 4.09 [3.59 to 4.67] | 1.52 [1.33 to 1.74]
  Flu B1 |  |  |  |  |  |  | 4.82 [3.66 to 6.34] | 6.85 [5.16 to 9.08] | 5.46 [4.06 to 7.35] | 5.40 [4.05 to 7.19] | 4.71 [3.56 to 6.23] | 6.14 [4.55 to 8.30] | 2.99 [2.23 to 4.00] | 3.54 [3.11 to 4.04] | 4.17 [3.67 to 4.75] | 4.57 [4.06 to 5.14] | 2.26 [2.00 to 2.55] | 3.05 [2.65 to 3.52] | 3.22 [2.81 to 3.70] | 4.00 [3.48 to 4.60] | 2.05 [1.79 to 2.36]
  Flu B2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 22 | 19 | 21 | 22 | 18 | 22 | 101 | 96 | 120 | 115 | 108 | 116 | 115 | 111
  Flu B2 |  |  |  |  |  |  | 4.82 [3.74 to 6.22] | 6.34 [4.87 to 8.25] | 6.04 [4.59 to 7.96] | 6.17 [4.73 to 8.05] | 4.91 [3.79 to 6.37] | 6.02 [4.53 to 8.00] | 2.68 [2.04 to 3.51] | 3.72 [3.33 to 4.16] | 4.16 [3.72 to 4.66] | 4.54 [4.10 to 5.02] | 1.81 [1.63 to 2.01] | 3.57 [3.19 to 4.00] | 3.83 [3.44 to 4.28] | 4.45 [3.99 to 4.97] | 2.10 [1.88 to 2.35]

16. Primary Outcome: Percentage of Participants With Antigen 2 Antibody SCR
Time Frame: From Day 1 to Day 29
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Flu mRNA_Ph1_1 Younger Adults (YA) Group | Flu mRNA_Ph1_2 YA Group | Flu mRNA_Ph1_3 YA Group | Flu mRNA_Ph1_4 YA Group | Flu mRNA_Ph1_5 YA Group | Flu mRNA_Ph1_6 YA Group | Flu mRNA_Ph1_7 YA Group | Flu mRNA_Ph1_8 YA Group | Flu mRNA_Ph1_9 YA Group | Flu mRNA_Ph1_10 YA Group | Flu mRNA_Ph1_11 YA Group | Flu mRNA_Ph1_12 YA Group | Control Ph1_YA Group | Flu mRNA_Ph2_1_YA Group | Flu mRNA_Ph2_2_YA Group | Flu mRNA_Ph2_3_YA Group | Control_Ph2_YA Group | Flu mRNA_Ph2_1_Older Adults (OA) Group | Flu mRNA_Ph2_2_OA Group | Flu mRNA_Ph2_3_OA Group | Control_Ph2_OA Group
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 22 | 19 | 21 | 22 | 19 | 22 | 101 | 97 | 121 | 115 | 108 | 116 | 115 | 111
Percentage of participants
  Flu A1 |  |  |  |  |  |  | 73.9 [51.6 to 89.8] | 63.6 [40.7 to 82.8] | 63.2 [38.4 to 83.7] | 76.2 [52.8 to 91.8] | 86.4 [65.1 to 97.1] | 78.9 [54.4 to 93.9] | 9.1 [1.1 to 29.2] | 68.3 [58.3 to 77.2] | 77.3 [67.7 to 85.2] | 77.7 [69.2 to 84.8] | 3.5 [1.0 to 8.7] | 58.3 [48.5 to 67.7] | 61.2 [51.7 to 70.1] | 72.2 [63.0 to 80.1] | 5.4 [2.0 to 11.4]
  Flu A2 |  |  |  |  |  |  | 39.1 [19.7 to 61.5] | 50.0 [28.2 to 71.8] | 52.6 [28.9 to 75.6] | 66.7 [43.0 to 85.4] | 54.5 [32.2 to 75.6] | 63.2 [38.4 to 83.7] | 18.2 [5.2 to 40.3] | 32.7 [23.7 to 42.7] | 46.4 [36.2 to 56.8] | 50.4 [41.2 to 59.6] | 7.0 [3.1 to 13.2] | 38.9 [29.7 to 48.7] | 40.5 [31.5 to 50.0] | 45.2 [35.9 to 54.8] | 6.3 [2.6 to 12.6]
  Flu B1 |  |  |  |  |  |  | 69.6 [47.1 to 86.8] | 77.3 [54.6 to 92.2] | 57.9 [33.5 to 79.7] | 57.1 [34.0 to 78.2] | 54.5 [32.2 to 75.6] | 63.2 [38.4 to 83.7] | 45.5 [24.4 to 67.8] | 38.6 [29.1 to 48.8] | 50.5 [40.2 to 60.8] | 61.2 [51.9 to 69.9] | 24.3 [16.8 to 33.2] | 39.8 [30.5 to 49.7] | 35.3 [26.7 to 44.8] | 48.7 [39.3 to 58.2] | 18.9 [12.1 to 27.5]
  Flu B2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 22 | 19 | 21 | 22 | 18 | 22 | 101 | 96 | 120 | 115 | 108 | 116 | 115 | 111
  Flu B2 |  |  |  |  |  |  | 69.6 [47.1 to 86.8] | 63.6 [40.7 to 82.8] | 57.9 [33.5 to 79.7] | 61.9 [38.4 to 81.9] | 54.5 [32.2 to 75.6] | 61.1 [35.7 to 82.7] | 27.3 [10.7 to 50.2] | 43.6 [33.7 to 53.8] | 49.0 [38.6 to 59.4] | 58.3 [49.0 to 67.3] | 5.2 [1.9 to 11.0] | 34.3 [25.4 to 44.0] | 44.8 [35.6 to 54.3] | 51.3 [41.8 to 60.7] | 13.5 [7.8 to 21.3]

17. Secondary Outcome: GMT of Antigen 1 Antibody Titer
Description: Assay 1= with egg propagated Influenza virus and Assay 2= with cell propagated Influenza virus.
Time Frame: At Day 92
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Flu mRNA_Ph1_1 Younger Adults (YA) Group | Flu mRNA_Ph1_2 YA Group | Flu mRNA_Ph1_3 YA Group | Flu mRNA_Ph1_4 YA Group | Flu mRNA_Ph1_5 YA Group | Flu mRNA_Ph1_6 YA Group | Flu mRNA_Ph1_7 YA Group | Flu mRNA_Ph1_8 YA Group | Flu mRNA_Ph1_9 YA Group | Flu mRNA_Ph1_10 YA Group | Flu mRNA_Ph1_11 YA Group | Flu mRNA_Ph1_12 YA Group | Control Ph1_YA Group | Flu mRNA_Ph2_1_YA Group | Flu mRNA_Ph2_2_YA Group | Flu mRNA_Ph2_3_YA Group | Control_Ph2_YA Group | Flu mRNA_Ph2_1_Older Adults (OA) Group | Flu mRNA_Ph2_2_OA Group | Flu mRNA_Ph2_3_OA Group | Control_Ph2_OA Group
Number analyzed (Participants) | 20 | 22 | 20 | 21 | 20 | 20 | 21 | 20 | 20 | 20 | 22 | 21 | 20 | 96 | 89 | 117 | 112 | 105 | 110 | 111 | 109
Titers
  Flu A1 Assay 1: number analyzed (Participants) | 20 | 22 | 20 | 21 | 20 | 20 | 21 | 20 | 20 | 20 | 22 | 21 | 20 | 96 | 86 | 115 | 111 | 105 | 107 | 108 | 109
  Flu A1 Assay 1 | 249.15 [173.16 to 358.51] | 192.79 [137.06 to 271.19] | 141.86 [99.24 to 202.76] | 170.29 [120.34 to 240.99] | 180.99 [126.21 to 259.54] | 161.89 [113.44 to 231.04] | 162.26 [114.31 to 230.34] | 181.10 [126.57 to 259.12] | 189.92 [133.06 to 271.09] | 186.49 [130.23 to 267.06] | 139.19 [98.69 to 196.29] | 157.89 [111.25 to 224.09] | 175.06 [121.70 to 251.82] | 35.51 [28.05 to 44.94] | 42.16 [33.07 to 53.73] | 49.93 [40.30 to 61.86] | 32.01 [25.76 to 39.78] | 45.30 [35.89 to 57.19] | 56.56 [44.85 to 71.32] | 54.03 [42.88 to 68.08] | 37.38 [29.75 to 46.96]
  Flu A2 Assay 1 | 11.75 [8.22 to 16.80] | 55.13 [39.43 to 77.07] | 29.95 [21.10 to 42.51] | 54.66 [38.86 to 76.87] | 29.31 [20.58 to 41.75] | 60.28 [42.50 to 85.51] | 39.46 [28.02 to 55.57] | 44.27 [31.12 to 62.96] | 43.27 [30.52 to 61.35] | 40.37 [28.34 to 57.49] | 55.76 [39.85 to 78.03] | 36.29 [25.74 to 51.18] | 18.15 [12.71 to 25.93] | 64.25 [52.60 to 78.47] | 71.59 [58.44 to 87.71] | 83.99 [70.12 to 100.61] | 39.61 [32.95 to 47.61] | 102.19 [83.56 to 124.97] | 106.65 [87.44 to 130.09] | 113.92 [93.61 to 138.65] | 71.02 [58.29 to 86.54]
  Flu B1 Assay 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 96 | 89 | 117 | 112 | 105 | 110 | 111 | 109
  Flu B1 Assay 1 |  |  |  |  |  |  |  |  |  |  |  |  |  | 357.44 [312.20 to 409.25] | 370.02 [322.42 to 424.65] | 399.21 [353.18 to 451.22] | 455.96 [402.50 to 516.53] | 522.16 [463.42 to 588.34] | 506.16 [450.05 to 569.26] | 521.79 [464.51 to 586.13] | 710.33 [631.89 to 798.49]
  Flu B1 Assay 2: number analyzed (Participants) | 20 | 22 | 20 | 21 | 20 | 20 | 21 | 20 | 20 | 20 | 22 | 20 | 19 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Flu B1 Assay 2 | 103.58 [81.09 to 132.31] | 181.64 [144.48 to 228.36] | 166.80 [131.32 to 211.86] | 190.14 [150.62 to 240.03] | 205.33 [160.99 to 261.88] | 159.14 [125.44 to 201.90] | 155.71 [123.25 to 196.74] | 200.39 [157.48 to 254.99] | 187.72 [147.77 to 238.47] | 178.11 [139.79 to 226.92] | 204.04 [162.18 to 256.71] | 184.58 [144.99 to 234.99] | 282.65 [219.83 to 363.40] |  |  |  |  |  |  |  |
  Flu B2 Assay 1: number analyzed (Participants) | 20 | 22 | 20 | 21 | 20 | 20 | 21 | 20 | 20 | 20 | 22 | 21 | 20 | 96 | 88 | 117 | 112 | 105 | 110 | 111 | 109
  Flu B2 Assay 1 | 219.10 [169.39 to 283.39] | 502.03 [394.47 to 638.93] | 383.24 [297.89 to 493.04] | 467.42 [365.66 to 597.49] | 537.37 [416.59 to 693.16] | 463.98 [361.11 to 596.16] | 405.98 [317.33 to 519.40] | 544.86 [423.01 to 701.82] | 486.21 [377.94 to 625.49] | 441.71 [342.34 to 569.94] | 446.45 [350.33 to 568.95] | 442.34 [345.41 to 566.47] | 722.16 [558.36 to 934.02] | 480.70 [413.79 to 558.42] | 520.76 [446.98 to 606.72] | 571.84 [499.62 to 654.49] | 716.31 [624.19 to 822.04] | 440.05 [388.12 to 498.93] | 473.09 [417.80 to 535.69] | 499.32 [441.83 to 564.29] | 599.30 [529.97 to 677.69]

18. Secondary Outcome: GMT of Antigen 1 Antibody Titer
Description: Assay 1= with egg propagated Influenza virus and Assay 2= with cell propagated Influenza virus.
Time Frame: At Day 183
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Flu mRNA_Ph1_1 Younger Adults (YA) Group | Flu mRNA_Ph1_2 YA Group | Flu mRNA_Ph1_3 YA Group | Flu mRNA_Ph1_4 YA Group | Flu mRNA_Ph1_5 YA Group | Flu mRNA_Ph1_6 YA Group | Flu mRNA_Ph1_7 YA Group | Flu mRNA_Ph1_8 YA Group | Flu mRNA_Ph1_9 YA Group | Flu mRNA_Ph1_10 YA Group | Flu mRNA_Ph1_11 YA Group | Flu mRNA_Ph1_12 YA Group | Control Ph1_YA Group | Flu mRNA_Ph2_1_YA Group | Flu mRNA_Ph2_2_YA Group | Flu mRNA_Ph2_3_YA Group | Control_Ph2_YA Group | Flu mRNA_Ph2_1_Older Adults (OA) Group | Flu mRNA_Ph2_2_OA Group | Flu mRNA_Ph2_3_OA Group | Control_Ph2_OA Group
Number analyzed (Participants) | 18 | 15 | 15 | 20 | 17 | 16 | 15 | 15 | 20 | 17 | 20 | 18 | 15 | 96 | 95 | 120 | 113 | 103 | 110 | 112 | 113
Titers
  Flu A1 Assay 1: number analyzed (Participants) | 17 | 15 | 15 | 20 | 17 | 16 | 15 | 15 | 20 | 17 | 20 | 18 | 15 | 95 | 92 | 117 | 112 | 103 | 108 | 108 | 113
  Flu A1 Assay 1 | 124.39 [82.01 to 188.69] | 118.75 [76.74 to 183.77] | 100.46 [64.59 to 156.25] | 98.64 [67.52 to 144.10] | 134.12 [88.53 to 203.19] | 96.19 [62.97 to 146.94] | 95.13 [61.04 to 148.27] | 104.62 [67.08 to 163.16] | 100.95 [69.06 to 147.57] | 81.46 [53.74 to 123.48] | 70.62 [48.02 to 103.85] | 81.54 [54.55 to 121.88] | 114.27 [73.07 to 178.71] | 25.63 [20.61 to 31.87] | 30.42 [24.42 to 37.90] | 34.40 [28.16 to 42.03] | 24.34 [19.90 to 29.77] | 30.51 [24.37 to 38.21] | 38.15 [30.59 to 47.58] | 40.80 [32.71 to 50.90] | 28.27 [22.79 to 35.06]
  Flu A2 Assay 1 | 12.27 [8.51 to 17.70] | 40.48 [27.31 to 60.01] | 20.58 [13.87 to 30.55] | 28.67 [20.36 to 40.36] | 20.24 [13.92 to 29.44] | 39.35 [26.84 to 57.71] | 23.54 [15.85 to 34.97] | 34.09 [22.84 to 50.89] | 31.34 [22.27 to 44.12] | 29.18 [20.02 to 42.53] | 29.37 [20.79 to 41.50] | 25.72 [17.89 to 36.97] | 12.73 [8.50 to 19.06] | 40.76 [33.62 to 49.42] | 46.04 [37.98 to 55.82] | 45.33 [38.02 to 54.04] | 30.65 [25.64 to 36.64] | 58.66 [48.07 to 71.59] | 66.14 [54.44 to 80.35] | 65.11 [53.72 to 78.92] | 44.85 [37.05 to 54.29]
  Flu B1 Assay 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 96 | 95 | 120 | 113 | 103 | 110 | 112 | 113
  Flu B1 Assay 1 |  |  |  |  |  |  |  |  |  |  |  |  |  | 315.92 [280.31 to 356.04] | 349.33 [309.97 to 393.68] | 338.71 [303.64 to 377.84] | 403.07 [360.83 to 450.26] | 453.91 [405.18 to 508.51] | 425.18 [380.53 to 475.08] | 469.87 [421.04 to 524.36] | 557.86 [500.33 to 622.00]
  Flu B1 Assay 2: number analyzed (Participants) | 18 | 15 | 15 | 20 | 17 | 16 | 15 | 15 | 20 | 17 | 20 | 17 | 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Flu B1 Assay 2 | 121.95 [93.94 to 158.30] | 159.09 [120.22 to 210.51] | 154.88 [117.10 to 204.85] | 165.36 [129.73 to 210.77] | 142.31 [108.80 to 186.16] | 146.00 [111.32 to 191.48] | 161.31 [121.84 to 213.56] | 208.89 [157.25 to 277.48] | 166.40 [130.45 to 212.26] | 196.59 [150.49 to 256.81] | 163.74 [128.14 to 209.21] | 171.47 [131.44 to 223.70] | 210.29 [156.09 to 283.32] |  |  |  |  |  |  |  |
  Flu B2 Assay 1: number analyzed (Participants) | 18 | 15 | 15 | 20 | 17 | 16 | 15 | 15 | 20 | 17 | 20 | 18 | 15 | 96 | 94 | 120 | 113 | 103 | 109 | 112 | 113
  Flu B2 Assay 1 | 290.27 [222.31 to 379.00] | 517.33 [388.49 to 688.89] | 444.01 [333.25 to 591.58] | 451.08 [351.73 to 578.49] | 498.91 [379.85 to 655.28] | 449.90 [340.69 to 594.12] | 413.03 [309.73 to 550.79] | 666.47 [498.26 to 891.47] | 489.90 [381.71 to 628.75] | 448.11 [340.62 to 589.53] | 461.80 [358.83 to 594.32] | 428.52 [329.05 to 558.08] | 791.84 [590.49 to 1061.84] | 350.40 [309.39 to 396.84] | 416.09 [367.34 to 471.31] | 424.47 [379.08 to 475.29] | 468.00 [417.20 to 525.00] | 291.02 [260.27 to 325.40] | 328.26 [294.08 to 366.41] | 340.46 [305.71 to 379.16] | 397.29 [357.09 to 442.01]

19. Secondary Outcome: GMI of Antigen 1 Antibody Titer From Day 1 to Day 92
Description: Assay 1= with egg propagated Influenza virus and Assay 2= with cell propagated Influenza virus.
Time Frame: From Day 1 (baseline) to Day 92
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Flu mRNA_Ph1_1 Younger Adults (YA) Group | Flu mRNA_Ph1_2 YA Group | Flu mRNA_Ph1_3 YA Group | Flu mRNA_Ph1_4 YA Group | Flu mRNA_Ph1_5 YA Group | Flu mRNA_Ph1_6 YA Group | Flu mRNA_Ph1_7 YA Group | Flu mRNA_Ph1_8 YA Group | Flu mRNA_Ph1_9 YA Group | Flu mRNA_Ph1_10 YA Group | Flu mRNA_Ph1_11 YA Group | Flu mRNA_Ph1_12 YA Group | Control Ph1_YA Group | Flu mRNA_Ph2_1_YA Group | Flu mRNA_Ph2_2_YA Group | Flu mRNA_Ph2_3_YA Group | Control_Ph2_YA Group | Flu mRNA_Ph2_1_Older Adults (OA) Group | Flu mRNA_Ph2_2_OA Group | Flu mRNA_Ph2_3_OA Group | Control_Ph2_OA Group
Number analyzed (Participants) | 20 | 22 | 20 | 21 | 20 | 20 | 21 | 20 | 20 | 20 | 22 | 21 | 20 | 96 | 89 | 117 | 112 | 105 | 110 | 111 | 109
Ratio
  Flu A1 Assay 1: number analyzed (Participants) | 20 | 22 | 20 | 21 | 20 | 20 | 21 | 20 | 20 | 20 | 22 | 21 | 20 | 96 | 86 | 115 | 111 | 105 | 107 | 108 | 109
  Flu A1 Assay 1 | 6.95 [4.83 to 10.00] | 5.38 [3.82 to 7.56] | 3.96 [2.77 to 5.66] | 4.75 [3.36 to 6.72] | 5.05 [3.52 to 7.24] | 4.52 [3.16 to 6.44] | 4.53 [3.19 to 6.42] | 5.05 [3.53 to 7.23] | 5.30 [3.71 to 7.56] | 5.20 [3.63 to 7.45] | 3.88 [2.75 to 5.48] | 4.40 [3.10 to 6.25] | 4.88 [3.39 to 7.02] | 4.58 [3.62 to 5.80] | 5.44 [4.27 to 6.93] | 6.44 [5.20 to 7.98] | 4.13 [3.32 to 5.13] | 4.85 [3.84 to 6.12] | 6.05 [4.80 to 7.63] | 5.78 [4.59 to 7.28] | 4.00 [3.18 to 5.02]
  Flu A2 Assay 1 | 1.00 [0.70 to 1.43] | 4.68 [3.35 to 6.54] | 2.54 [1.79 to 3.61] | 4.64 [3.30 to 6.52] | 2.49 [1.75 to 3.54] | 5.11 [3.61 to 7.25] | 3.35 [2.38 to 4.71] | 3.76 [2.64 to 5.34] | 3.67 [2.59 to 5.20] | 3.42 [2.40 to 4.88] | 4.73 [3.38 to 6.62] | 3.08 [2.18 to 4.34] | 1.54 [1.08 to 2.20] | 4.57 [3.74 to 5.59] | 5.10 [4.16 to 6.24] | 5.98 [4.99 to 7.16] | 2.82 [2.35 to 3.39] | 5.42 [4.43 to 6.63] | 5.66 [4.64 to 6.90] | 6.05 [4.97 to 7.36] | 3.77 [3.09 to 4.59]
  Flu B1 Assay 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 96 | 89 | 117 | 112 | 105 | 110 | 111 | 109
  Flu B1 Assay 1 |  |  |  |  |  |  |  |  |  |  |  |  |  | 1.81 [1.58 to 2.07] | 1.87 [1.63 to 2.15] | 2.02 [1.78 to 2.28] | 2.30 [2.03 to 2.61] | 2.35 [2.09 to 2.65] | 2.28 [2.03 to 2.56] | 2.35 [2.09 to 2.64] | 3.20 [2.84 to 3.59]
  Flu B1 Assay 2: number analyzed (Participants) | 20 | 22 | 20 | 21 | 20 | 20 | 21 | 20 | 20 | 20 | 22 | 20 | 19 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Flu B1 Assay 2 | 1.27 [0.99 to 1.62] | 2.23 [1.77 to 2.80] | 2.05 [1.61 to 2.60] | 2.33 [1.85 to 2.94] | 2.52 [1.97 to 3.21] | 1.95 [1.54 to 2.48] | 1.91 [1.51 to 2.41] | 2.46 [1.93 to 3.13] | 2.30 [1.81 to 2.92] | 2.18 [1.71 to 2.78] | 2.50 [1.99 to 3.15] | 2.26 [1.78 to 2.88] | 3.47 [2.70 to 4.46] |  |  |  |  |  |  |  |
  Flu B2 Assay 1: number analyzed (Participants) | 20 | 22 | 20 | 21 | 20 | 20 | 21 | 20 | 20 | 20 | 22 | 21 | 20 | 96 | 88 | 117 | 112 | 105 | 110 | 111 | 109
  Flu B2 Assay 1 | 0.98 [0.76 to 1.27] | 2.25 [1.77 to 2.86] | 1.72 [1.33 to 2.21] | 2.09 [1.64 to 2.67] | 2.41 [1.86 to 3.10] | 2.08 [1.62 to 2.67] | 1.82 [1.42 to 2.33] | 2.44 [1.89 to 3.14] | 2.18 [1.69 to 2.80] | 1.98 [1.53 to 2.55] | 2.00 [1.57 to 2.55] | 1.98 [1.55 to 2.54] | 3.23 [2.50 to 4.18] | 1.63 [1.41 to 1.90] | 1.77 [1.52 to 2.06] | 1.94 [1.70 to 2.22] | 2.43 [2.12 to 2.79] | 2.05 [1.81 to 2.33] | 2.21 [1.95 to 2.50] | 2.33 [2.06 to 2.63] | 2.80 [2.47 to 3.16]

20. Secondary Outcome: GMI of Antigen 1 Antibody Titer From Day 1 to Day 183
Description: Assay 1= with egg propagated Influenza virus and Assay 2= with cell propagated Influenza virus.
Time Frame: From Day 1 (baseline) to Day 183
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Flu mRNA_Ph1_1 Younger Adults (YA) Group | Flu mRNA_Ph1_2 YA Group | Flu mRNA_Ph1_3 YA Group | Flu mRNA_Ph1_4 YA Group | Flu mRNA_Ph1_5 YA Group | Flu mRNA_Ph1_6 YA Group | Flu mRNA_Ph1_7 YA Group | Flu mRNA_Ph1_8 YA Group | Flu mRNA_Ph1_9 YA Group | Flu mRNA_Ph1_10 YA Group | Flu mRNA_Ph1_11 YA Group | Flu mRNA_Ph1_12 YA Group | Control Ph1_YA Group | Flu mRNA_Ph2_1_YA Group | Flu mRNA_Ph2_2_YA Group | Flu mRNA_Ph2_3_YA Group | Control_Ph2_YA Group | Flu mRNA_Ph2_1_Older Adults (OA) Group | Flu mRNA_Ph2_2_OA Group | Flu mRNA_Ph2_3_OA Group | Control_Ph2_OA Group
Number analyzed (Participants) | 18 | 15 | 15 | 20 | 17 | 16 | 15 | 15 | 20 | 17 | 20 | 18 | 15 | 96 | 95 | 120 | 113 | 103 | 110 | 112 | 113
Ratio
  Flu A1 Assay 1: number analyzed (Participants) | 17 | 15 | 15 | 20 | 17 | 16 | 15 | 15 | 20 | 17 | 20 | 18 | 15 | 95 | 92 | 117 | 112 | 103 | 108 | 108 | 113
  Flu A1 Assay 1 | 3.55 [2.34 to 5.39] | 3.39 [2.19 to 5.25] | 2.87 [1.84 to 4.46] | 2.82 [1.93 to 4.11] | 3.83 [2.53 to 5.80] | 2.75 [1.80 to 4.20] | 2.72 [1.74 to 4.23] | 2.99 [1.92 to 4.66] | 2.88 [1.97 to 4.21] | 2.33 [1.53 to 3.53] | 2.02 [1.37 to 2.97] | 2.33 [1.56 to 3.48] | 3.26 [2.09 to 5.10] | 3.23 [2.60 to 4.02] | 3.84 [3.08 to 4.78] | 4.34 [3.55 to 5.30] | 3.07 [2.51 to 3.76] | 3.20 [2.55 to 4.01] | 4.00 [3.21 to 4.99] | 4.28 [3.43 to 5.34] | 2.96 [2.39 to 3.68]
  Flu A2 Assay 1 | 1.06 [0.73 to 1.53] | 3.49 [2.35 to 5.17] | 1.77 [1.20 to 2.63] | 2.47 [1.76 to 3.48] | 1.74 [1.20 to 2.54] | 3.39 [2.31 to 4.97] | 2.03 [1.37 to 3.01] | 2.94 [1.97 to 4.39] | 2.70 [1.92 to 3.80] | 2.51 [1.73 to 3.67] | 2.53 [1.79 to 3.58] | 2.22 [1.54 to 3.19] | 1.10 [0.73 to 1.64] | 2.85 [2.35 to 3.46] | 3.22 [2.66 to 3.91] | 3.17 [2.66 to 3.78] | 2.15 [1.79 to 2.57] | 2.99 [2.45 to 3.65] | 3.37 [2.78 to 4.10] | 3.32 [2.74 to 4.03] | 2.29 [1.89 to 2.77]
  Flu B1 Assay 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 96 | 95 | 120 | 113 | 103 | 110 | 112 | 113
  Flu B1 Assay 1 |  |  |  |  |  |  |  |  |  |  |  |  |  | 1.58 [1.41 to 1.79] | 1.75 [1.56 to 1.97] | 1.70 [1.52 to 1.90] | 2.02 [1.81 to 2.26] | 2.02 [1.81 to 2.27] | 1.89 [1.70 to 2.12] | 2.09 [1.88 to 2.34] | 2.49 [2.23 to 2.77]
  Flu B1 Assay 2: number analyzed (Participants) | 18 | 15 | 15 | 20 | 17 | 16 | 15 | 15 | 20 | 17 | 20 | 17 | 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Flu B1 Assay 2 | 1.50 [1.16 to 1.95] | 1.96 [1.48 to 2.59] | 1.91 [1.44 to 2.52] | 2.04 [1.60 to 2.60] | 1.75 [1.34 to 2.29] | 1.80 [1.37 to 2.36] | 1.99 [1.50 to 2.63] | 2.57 [1.94 to 3.42] | 2.05 [1.61 to 2.61] | 2.42 [1.85 to 3.16] | 2.02 [1.58 to 2.58] | 2.11 [1.62 to 2.75] | 2.59 [1.92 to 3.49] |  |  |  |  |  |  |  |
  Flu B2 Assay 1: number analyzed (Participants) | 18 | 15 | 15 | 20 | 17 | 16 | 15 | 15 | 20 | 17 | 20 | 18 | 15 | 96 | 94 | 120 | 113 | 103 | 109 | 112 | 113
  Flu B2 Assay 1 | 1.31 [1.00 to 1.71] | 2.34 [1.75 to 3.11] | 2.01 [1.51 to 2.67] | 2.04 [1.59 to 2.61] | 2.25 [1.72 to 2.96] | 2.03 [1.54 to 2.68] | 1.87 [1.40 to 2.49] | 3.01 [2.25 to 4.03] | 2.21 [1.72 to 2.84] | 2.02 [1.54 to 2.66] | 2.09 [1.62 to 2.68] | 1.94 [1.49 to 2.52] | 3.58 [2.67 to 4.80] | 1.16 [1.03 to 1.32] | 1.38 [1.22 to 1.57] | 1.41 [1.26 to 1.58] | 1.56 [1.39 to 1.74] | 1.34 [1.19 to 1.49] | 1.51 [1.35 to 1.68] | 1.56 [1.40 to 1.74] | 1.82 [1.64 to 2.03]

21. Secondary Outcome: Percentage of Participants With Antigen 1 Antibody SPR
Description: Assay 1= with egg propagated Influenza virus and Assay 2= with cell propagated Influenza virus.
Time Frame: At Day 183
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Flu mRNA_Ph1_1 Younger Adults (YA) Group | Flu mRNA_Ph1_2 YA Group | Flu mRNA_Ph1_3 YA Group | Flu mRNA_Ph1_4 YA Group | Flu mRNA_Ph1_5 YA Group | Flu mRNA_Ph1_6 YA Group | Flu mRNA_Ph1_7 YA Group | Flu mRNA_Ph1_8 YA Group | Flu mRNA_Ph1_9 YA Group | Flu mRNA_Ph1_10 YA Group | Flu mRNA_Ph1_11 YA Group | Flu mRNA_Ph1_12 YA Group | Control Ph1_YA Group | Flu mRNA_Ph2_1_YA Group | Flu mRNA_Ph2_2_YA Group | Flu mRNA_Ph2_3_YA Group | Control_Ph2_YA Group | Flu mRNA_Ph2_1_Older Adults (OA) Group | Flu mRNA_Ph2_2_OA Group | Flu mRNA_Ph2_3_OA Group | Control_Ph2_OA Group
Number analyzed (Participants) | 18 | 15 | 15 | 20 | 17 | 16 | 15 | 15 | 20 | 17 | 20 | 18 | 15 | 96 | 95 | 120 | 113 | 103 | 110 | 112 | 113
Percentage of participants
  Flu A1 Assay 1: number analyzed (Participants) | 17 | 15 | 15 | 20 | 17 | 16 | 15 | 15 | 20 | 17 | 20 | 18 | 15 | 95 | 95 | 118 | 113 | 103 | 108 | 110 | 113
  Flu A1 Assay 1 | 94.1 [71.3 to 99.9] | 93.3 [68.1 to 99.8] | 86.7 [59.5 to 98.3] | 95.0 [75.1 to 99.9] | 100 [80.5 to 100] | 81.3 [54.4 to 96.0] | 93.3 [68.1 to 99.8] | 80.0 [51.9 to 95.7] | 95.0 [75.1 to 99.9] | 82.4 [56.6 to 96.2] | 65.0 [40.8 to 84.6] | 77.8 [52.4 to 93.6] | 86.7 [59.5 to 98.3] | 44.2 [34.0 to 54.8] | 47.4 [37.0 to 57.9] | 47.5 [38.2 to 56.9] | 37.2 [28.3 to 46.8] | 39.8 [30.3 to 49.9] | 48.1 [38.4 to 58.0] | 51.8 [42.1 to 61.4] | 40.7 [31.6 to 50.4]
  Flu A2 Assay 1 | 22.2 [6.4 to 47.6] | 66.7 [38.4 to 88.2] | 46.7 [21.3 to 73.4] | 60.0 [36.1 to 80.9] | 47.1 [23.0 to 72.2] | 56.3 [29.9 to 80.2] | 46.7 [21.3 to 73.4] | 73.3 [44.9 to 92.2] | 50.0 [27.2 to 72.8] | 52.9 [27.8 to 77.0] | 45.0 [23.1 to 68.5] | 50.0 [26.0 to 74.0] | 33.3 [11.8 to 61.6] | 59.4 [48.9 to 69.3] | 63.2 [52.6 to 72.8] | 64.2 [54.9 to 72.7] | 54.9 [45.2 to 64.2] | 67.0 [57.0 to 75.9] | 66.4 [56.7 to 75.1] | 70.5 [61.2 to 78.8] | 58.4 [48.8 to 67.6]
  Flu B1 Assay 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 96 | 95 | 120 | 113 | 103 | 110 | 112 | 113
  Flu B1 Assay 1 |  |  |  |  |  |  |  |  |  |  |  |  |  | 100 [96.2 to 100] | 100 [96.2 to 100] | 100 [97.0 to 100] | 100 [96.8 to 100] | 100 [96.5 to 100] | 100 [96.7 to 100] | 100 [96.8 to 100] | 100 [96.8 to 100]
  Flu B1 Assay 2: number analyzed (Participants) | 18 | 15 | 15 | 20 | 17 | 16 | 15 | 15 | 20 | 17 | 20 | 18 | 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Flu B1 Assay 2 | 88.9 [65.3 to 98.6] | 100 [78.2 to 100] | 100 [78.2 to 100] | 100 [83.2 to 100] | 100 [80.5 to 100] | 100 [79.4 to 100] | 100 [78.2 to 100] | 100 [78.2 to 100] | 100 [83.2 to 100] | 100 [80.5 to 100] | 100 [83.2 to 100] | 100 [81.5 to 100] | 100 [78.2 to 100] |  |  |  |  |  |  |  |
  Flu B2 Assay 1: number analyzed (Participants) | 18 | 15 | 15 | 20 | 17 | 16 | 15 | 15 | 20 | 17 | 20 | 18 | 15 | 96 | 95 | 120 | 113 | 103 | 109 | 112 | 113
  Flu B2 Assay 1 | 100 [81.5 to 100] | 100 [78.2 to 100] | 100 [78.2 to 100] | 100 [83.2 to 100] | 100 [80.5 to 100] | 100 [79.4 to 100] | 100 [78.2 to 100] | 100 [78.2 to 100] | 100 [83.2 to 100] | 100 [80.5 to 100] | 100 [83.2 to 100] | 100 [81.5 to 100] | 100 [78.2 to 100] | 100 [96.2 to 100] | 100 [96.2 to 100] | 100 [97.0 to 100] | 100 [96.8 to 100] | 99.0 [94.7 to 100] | 100 [96.7 to 100] | 100 [96.8 to 100] | 100 [96.8 to 100]

22. Secondary Outcome: GMT of Antigen 2 Antibody Titer
Time Frame: At Day 92 and Day 183
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Flu mRNA_Ph1_1 Younger Adults (YA) Group | Flu mRNA_Ph1_2 YA Group | Flu mRNA_Ph1_3 YA Group | Flu mRNA_Ph1_4 YA Group | Flu mRNA_Ph1_5 YA Group | Flu mRNA_Ph1_6 YA Group | Flu mRNA_Ph1_7 YA Group | Flu mRNA_Ph1_8 YA Group | Flu mRNA_Ph1_9 YA Group | Flu mRNA_Ph1_10 YA Group | Flu mRNA_Ph1_11 YA Group | Flu mRNA_Ph1_12 YA Group | Control Ph1_YA Group | Flu mRNA_Ph2_1_YA Group | Flu mRNA_Ph2_2_YA Group | Flu mRNA_Ph2_3_YA Group | Control_Ph2_YA Group | Flu mRNA_Ph2_1_Older Adults (OA) Group | Flu mRNA_Ph2_2_OA Group | Flu mRNA_Ph2_3_OA Group | Control_Ph2_OA Group
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 20 | 20 | 20 | 22 | 21 | 20 | 96 | 95 | 120 | 113 | 105 | 110 | 112 | 113
Titers
  Flu A1, Post-dosing at Day 92: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 20 | 20 | 20 | 22 | 21 | 20 | 96 | 89 | 117 | 112 | 105 | 110 | 111 | 108
  Flu A1, Post-dosing at Day 92 |  |  |  |  |  |  | 3413.56 [2608.88 to 4466.45] | 3012.57 [2280.43 to 3979.78] | 2965.07 [2254.80 to 3899.08] | 3738.95 [2826.14 to 4946.58] | 3441.57 [2638.90 to 4488.39] | 4274.50 [3261.91 to 5601.42] | 1169.80 [877.58 to 1559.32] | 571.40 [478.17 to 682.80] | 722.85 [602.29 to 867.53] | 734.36 [624.97 to 862.91] | 128.40 [108.98 to 151.28] | 684.46 [583.38 to 803.06] | 674.07 [575.98 to 788.85] | 791.40 [677.27 to 924.77] | 172.46 [147.38 to 201.79]
  Flu A1, Post-dosing at Day 183: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 15 | 20 | 17 | 20 | 18 | 15 | 96 | 95 | 120 | 113 | 103 | 110 | 112 | 113
  Flu A1, Post-dosing at Day 183 |  |  |  |  |  |  | 3564.38 [2560.66 to 4961.53] | 2635.37 [1880.45 to 3693.34] | 2682.13 [2018.21 to 3564.44] | 3489.51 [2546.78 to 4781.21] | 3472.42 [2596.95 to 4643.03] | 4239.44 [3136.10 to 5730.94] | 1048.36 [741.30 to 1482.62] | 444.85 [370.47 to 534.16] | 534.28 [444.54 to 642.14] | 545.14 [461.18 to 644.39] | 132.78 [112.08 to 157.30] | 532.03 [446.15 to 634.43] | 470.78 [396.55 to 558.89] | 612.30 [516.57 to 725.78] | 166.23 [140.42 to 196.79]
  Flu A2, Post-dosing at Day 92: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 20 | 20 | 20 | 22 | 21 | 20 | 96 | 89 | 117 | 112 | 105 | 110 | 111 | 108
  Flu A2, Post-dosing at Day 92 |  |  |  |  |  |  | 637.45 [519.98 to 781.47] | 844.82 [683.69 to 1043.93] | 636.20 [517.35 to 782.37] | 696.15 [561.66 to 862.84] | 784.67 [641.72 to 959.47] | 844.05 [685.93 to 1038.61] | 411.14 [330.13 to 512.03] | 827.90 [734.62 to 933.03] | 875.59 [775.24 to 988.93] | 1005.14 [901.57 to 1120.61] | 416.04 [372.71 to 464.40] | 1202.72 [1070.36 to 1351.46] | 1275.88 [1137.26 to 1431.40] | 1394.04 [1244.06 to 1562.11] | 566.45 [505.00 to 635.39]
  Flu A2, Post-dosing at Day 183: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 15 | 20 | 17 | 20 | 18 | 15 | 96 | 95 | 120 | 113 | 103 | 110 | 112 | 113
  Flu A2, Post-dosing at Day 183 |  |  |  |  |  |  | 482.94 [365.04 to 638.93] | 691.16 [517.52 to 923.07] | 538.10 [422.45 to 685.42] | 593.16 [451.41 to 779.42] | 653.49 [510.58 to 836.39] | 661.58 [510.14 to 857.99] | 302.98 [225.20 to 407.64] | 492.09 [440.03 to 550.32] | 551.37 [492.98 to 616.68] | 585.21 [528.14 to 648.44] | 271.70 [244.99 to 301.31] | 727.45 [644.79 to 820.72] | 700.38 [622.60 to 787.88] | 816.15 [726.38 to 917.02] | 397.88 [354.41 to 446.67]
  Flu B1, Post-dosing at Day 92: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 20 | 20 | 20 | 22 | 21 | 20 | 96 | 89 | 117 | 112 | 105 | 110 | 111 | 108
  Flu B1, Post-dosing at Day 92 |  |  |  |  |  |  | 365.32 [275.53 to 484.38] | 576.79 [431.04 to 771.82] | 401.61 [301.39 to 535.16] | 483.67 [361.55 to 647.04] | 385.93 [292.19 to 509.74] | 438.90 [329.69 to 584.30] | 261.90 [193.56 to 354.37] | 409.51 [361.20 to 464.28] | 501.61 [441.78 to 569.55] | 512.92 [458.15 to 574.23] | 267.02 [237.93 to 299.66] | 538.58 [470.60 to 616.38] | 574.01 [502.80 to 655.30] | 611.15 [535.89 to 696.97] | 355.51 [311.44 to 405.82]
  Flu B1, Post-dosing at Day 183: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 15 | 20 | 17 | 20 | 18 | 15 | 96 | 95 | 120 | 113 | 103 | 110 | 112 | 113
  Flu B1, Post-dosing at Day 183 |  |  |  |  |  |  | 384.20 [276.74 to 533.38] | 716.17 [511.59 to 1002.56] | 439.50 [330.94 to 583.68] | 586.65 [429.01 to 802.23] | 419.67 [314.35 to 560.29] | 484.54 [357.96 to 655.88] | 326.16 [230.47 to 461.58] | 307.31 [272.34 to 346.78] | 371.76 [329.66 to 419.23] | 372.01 [333.35 to 415.16] | 221.57 [198.20 to 247.69] | 375.13 [332.23 to 423.57] | 388.81 [345.37 to 437.72] | 449.14 [399.38 to 505.10] | 288.98 [257.24 to 324.65]
  Flu B2, Post-dosing at Day 92: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 20 | 20 | 20 | 22 | 21 | 20 | 96 | 89 | 117 | 112 | 105 | 110 | 111 | 108
  Flu B2, Post-dosing at Day 92 |  |  |  |  |  |  | 1815.84 [1413.39 to 2332.89] | 2569.92 [1982.50 to 3331.39] | 1866.83 [1445.98 to 2410.18] | 2361.25 [1822.40 to 3059.42] | 1762.98 [1376.82 to 2257.45] | 1909.41 [1483.64 to 2457.36] | 1298.81 [992.67 to 1699.36] | 1966.97 [1784.99 to 2167.49] | 2217.80 [2008.88 to 2448.46] | 2214.84 [2028.65 to 2418.13] | 1080.66 [987.93 to 1182.10] | 2649.22 [2383.01 to 2945.16] | 2803.91 [2525.91 to 3112.50] | 3061.97 [2760.37 to 3396.52] | 1725.34 [1554.32 to 1915.18]
  Flu B2, Post-dosing at Day 183: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 15 | 20 | 17 | 20 | 18 | 15 | 96 | 95 | 120 | 113 | 103 | 110 | 112 | 113
  Flu B2, Post-dosing at Day 183 |  |  |  |  |  |  | 1633.79 [1240.95 to 2150.98] | 2310.02 [1742.83 to 3061.81] | 1613.52 [1271.80 to 2047.06] | 2262.11 [1739.52 to 2941.69] | 1513.91 [1188.47 to 1928.46] | 1744.56 [1356.31 to 2243.96] | 1187.10 [888.30 to 1586.40] | 1494.07 [1340.65 to 1665.05] | 1722.00 [1544.83 to 1919.48] | 1688.96 [1529.84 to 1864.62] | 940.94 [850.96 to 1040.42] | 1923.64 [1731.04 to 2137.67] | 2036.73 [1837.19 to 2257.94] | 2288.21 [2065.66 to 2534.74] | 1464.14 [1323.11 to 1620.21]

23. Secondary Outcome: GMI of Antigen 2 Antibody Titer
Time Frame: From Day 1 to Day 92 and Day 1 to Day 183
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Flu mRNA_Ph1_1 Younger Adults (YA) Group | Flu mRNA_Ph1_2 YA Group | Flu mRNA_Ph1_3 YA Group | Flu mRNA_Ph1_4 YA Group | Flu mRNA_Ph1_5 YA Group | Flu mRNA_Ph1_6 YA Group | Flu mRNA_Ph1_7 YA Group | Flu mRNA_Ph1_8 YA Group | Flu mRNA_Ph1_9 YA Group | Flu mRNA_Ph1_10 YA Group | Flu mRNA_Ph1_11 YA Group | Flu mRNA_Ph1_12 YA Group | Control Ph1_YA Group | Flu mRNA_Ph2_1_YA Group | Flu mRNA_Ph2_2_YA Group | Flu mRNA_Ph2_3_YA Group | Control_Ph2_YA Group | Flu mRNA_Ph2_1_Older Adults (OA) Group | Flu mRNA_Ph2_2_OA Group | Flu mRNA_Ph2_3_OA Group | Control_Ph2_OA Group
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 20 | 20 | 20 | 22 | 21 | 20 | 96 | 95 | 120 | 113 | 105 | 110 | 112 | 113
Ratio
  Flu A1, Post-dosing at Day 92: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 20 | 20 | 20 | 22 | 21 | 20 | 96 | 89 | 117 | 112 | 105 | 110 | 111 | 108
  Flu A1, Post-dosing at Day 92 |  |  |  |  |  |  | 4.24 [3.24 to 5.55] | 3.74 [2.83 to 4.94] | 3.68 [2.80 to 4.84] | 4.64 [3.51 to 6.14] | 4.27 [3.28 to 5.57] | 5.31 [4.05 to 6.95] | 1.45 [1.09 to 1.94] | 4.83 [4.04 to 5.77] | 6.11 [5.09 to 7.33] | 6.20 [5.28 to 7.29] | 1.08 [0.92 to 1.28] | 4.75 [4.05 to 5.57] | 4.67 [3.99 to 5.47] | 5.49 [4.70 to 6.41] | 1.20 [1.02 to 1.40]
  Flu A1, Post-dosing at Day 183: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 15 | 20 | 17 | 20 | 18 | 15 | 96 | 95 | 120 | 113 | 103 | 110 | 112 | 113
  Flu A1, Post-dosing at Day 183 |  |  |  |  |  |  | 4.19 [3.01 to 5.83] | 3.10 [2.21 to 4.34] | 3.15 [2.37 to 4.19] | 4.10 [2.99 to 5.62] | 4.08 [3.05 to 5.46] | 4.98 [3.69 to 6.74] | 1.23 [0.87 to 1.74] | 3.77 [3.14 to 4.53] | 4.53 [3.77 to 5.45] | 4.62 [3.91 to 5.47] | 1.13 [0.95 to 1.33] | 3.73 [3.13 to 4.45] | 3.30 [2.78 to 3.92] | 4.30 [3.62 to 5.09] | 1.17 [0.99 to 1.38]
  Flu A2, Post-dosing at Day 92: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 20 | 20 | 20 | 22 | 21 | 20 | 96 | 89 | 117 | 112 | 105 | 110 | 111 | 108
  Flu A2, Post-dosing at Day 92 |  |  |  |  |  |  | 3.28 [2.67 to 4.02] | 4.35 [3.52 to 5.37] | 3.27 [2.66 to 4.02] | 3.58 [2.89 to 4.44] | 4.04 [3.30 to 4.93] | 4.34 [3.53 to 5.34] | 2.11 [1.70 to 2.63] | 3.41 [3.03 to 3.84] | 3.61 [3.19 to 4.07] | 4.14 [3.71 to 4.62] | 1.71 [1.54 to 1.91] | 3.62 [3.22 to 4.07] | 3.84 [3.42 to 4.31] | 4.20 [3.75 to 4.70] | 1.71 [1.52 to 1.91]
  Flu A2, Post-dosing at Day 183: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 15 | 20 | 17 | 20 | 18 | 15 | 96 | 95 | 120 | 113 | 103 | 110 | 112 | 113
  Flu A2, Post-dosing at Day 183 |  |  |  |  |  |  | 2.54 [1.92 to 3.36] | 3.63 [2.72 to 4.85] | 2.83 [2.22 to 3.60] | 3.12 [2.37 to 4.09] | 3.43 [2.68 to 4.39] | 3.48 [2.68 to 4.51] | 1.59 [1.18 to 2.14] | 2.02 [1.81 to 2.26] | 2.26 [2.03 to 2.53] | 2.40 [2.17 to 2.66] | 1.12 [1.01 to 1.24] | 2.18 [1.94 to 2.46] | 2.10 [1.87 to 2.37] | 2.45 [2.18 to 2.75] | 1.19 [1.06 to 1.34]
  Flu B1, Post-dosing at Day 92: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 20 | 20 | 20 | 22 | 21 | 20 | 96 | 89 | 117 | 112 | 105 | 110 | 111 | 108
  Flu B1, Post-dosing at Day 92 |  |  |  |  |  |  | 1.23 [0.93 to 1.63] | 1.94 [1.45 to 2.59] | 1.35 [1.01 to 1.80] | 1.63 [1.22 to 2.18] | 1.30 [0.98 to 1.71] | 1.48 [1.11 to 1.96] | 0.88 [0.65 to 1.19] | 2.43 [2.15 to 2.76] | 2.98 [2.63 to 3.38] | 3.05 [2.72 to 3.41] | 1.59 [1.41 to 1.78] | 2.29 [2.00 to 2.62] | 2.44 [2.14 to 2.78] | 2.60 [2.28 to 2.96] | 1.51 [1.32 to 1.72]
  Flu B1, Post-dosing at Day 183: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 15 | 20 | 17 | 20 | 18 | 15 | 96 | 95 | 120 | 113 | 103 | 110 | 112 | 113
  Flu B1, Post-dosing at Day 183 |  |  |  |  |  |  | 1.27 [0.91 to 1.76] | 2.36 [1.69 to 3.31] | 1.45 [1.09 to 1.93] | 1.94 [1.42 to 2.65] | 1.39 [1.04 to 1.85] | 1.60 [1.18 to 2.16] | 1.08 [0.76 to 1.52] | 1.82 [1.61 to 2.05] | 2.20 [1.95 to 2.48] | 2.20 [1.97 to 2.46] | 1.31 [1.17 to 1.47] | 1.57 [1.39 to 1.78] | 1.63 [1.45 to 1.84] | 1.88 [1.68 to 2.12] | 1.21 [1.08 to 1.36]
  Flu B2, Post-dosing at Day 92: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 20 | 20 | 20 | 22 | 21 | 20 | 96 | 89 | 117 | 112 | 105 | 110 | 111 | 108
  Flu B2, Post-dosing at Day 92 |  |  |  |  |  |  | 3.46 [2.70 to 4.45] | 4.90 [3.78 to 6.35] | 3.56 [2.76 to 4.60] | 4.50 [3.48 to 5.83] | 3.36 [2.63 to 4.31] | 3.64 [2.83 to 4.69] | 2.48 [1.89 to 3.24] | 2.80 [2.54 to 3.08] | 3.15 [2.86 to 3.48] | 3.15 [2.88 to 3.44] | 1.54 [1.40 to 1.68] | 2.84 [2.55 to 3.15] | 3.00 [2.70 to 3.33] | 3.28 [2.95 to 3.63] | 1.85 [1.66 to 2.05]
  Flu B2, Post-dosing at Day 183: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 15 | 20 | 17 | 20 | 18 | 15 | 96 | 95 | 120 | 113 | 103 | 110 | 112 | 113
  Flu B2, Post-dosing at Day 183 |  |  |  |  |  |  | 3.05 [2.31 to 4.01] | 4.31 [3.25 to 5.71] | 3.01 [2.37 to 3.82] | 4.22 [3.24 to 5.49] | 2.82 [2.22 to 3.60] | 3.25 [2.53 to 4.18] | 2.21 [1.66 to 2.96] | 2.12 [1.90 to 2.36] | 2.44 [2.19 to 2.72] | 2.39 [2.17 to 2.64] | 1.33 [1.21 to 1.47] | 2.03 [1.82 to 2.25] | 2.15 [1.94 to 2.38] | 2.41 [2.18 to 2.67] | 1.54 [1.39 to 1.71]

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected from Day 1 to Day 7; Unsolicited AEs: Day 1 to day 28; All-cause mortality, SAEs, AESIs, and MAEs: from first vaccination (Day 1) up to study end (Day 183)
Arm/Group | Flu mRNA_Ph1_1 Younger Adults (YA) Group | Flu mRNA_Ph1_2 YA Group | Flu mRNA_Ph1_3 YA Group | Flu mRNA_Ph1_4 YA Group | Flu mRNA_Ph1_5 YA Group | Flu mRNA_Ph1_6 YA Group | Flu mRNA_Ph1_7 YA Group | Flu mRNA_Ph1_8 YA Group | Flu mRNA_Ph1_9 YA Group | Flu mRNA_Ph1_10 YA Group | Flu mRNA_Ph1_11 YA Group | Flu mRNA_Ph1_12 YA Group | Control Ph1_YA Group | Flu mRNA_Ph2_1_YA Group | Flu mRNA_Ph2_2_YA Group | Flu mRNA_Ph2_3_YA Group | Control_Ph2_YA Group | Flu mRNA_Ph2_1_Older Adults (OA) Group | Flu mRNA_Ph2_2_OA Group | Flu mRNA_Ph2_3_OA Group | Control_Ph2_OA Group
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/22 | 0/23 | 0/23 | 0/22 | 0/25 | 0/23 | 0/22 | 0/23 | 0/22 | 0/23 | 0/21 | 0/23 | 0/115 | 0/108 | 0/137 | 0/120 | 0/119 | 0/122 | 0/125 | 0/117
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22 | 0/23 | 0/23 | 0/22 | 1/25 | 0/23 | 0/22 | 0/23 | 0/22 | 0/23 | 1/21 | 0/23 | 0/115 | 1/108 | 0/137 | 3/120 | 3/119 | 6/122 | 2/125 | 2/117
Other Adverse Events (participants affected / at risk) | 16/21 | 22/22 | 23/23 | 22/23 | 20/22 | 24/25 | 22/23 | 20/22 | 19/23 | 20/22 | 23/23 | 19/21 | 18/23 | 99/115 | 95/108 | 127/137 | 89/120 | 83/119 | 88/122 | 91/125 | 69/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flu mRNA_Ph1_1 Younger Adults (YA) Group (N=21) | Flu mRNA_Ph1_2 YA Group (N=22) | Flu mRNA_Ph1_3 YA Group (N=23) | Flu mRNA_Ph1_4 YA Group (N=23) | Flu mRNA_Ph1_5 YA Group (N=22) | Flu mRNA_Ph1_6 YA Group (N=25) | Flu mRNA_Ph1_7 YA Group (N=23) | Flu mRNA_Ph1_8 YA Group (N=22) | Flu mRNA_Ph1_9 YA Group (N=23) | Flu mRNA_Ph1_10 YA Group (N=22) | Flu mRNA_Ph1_11 YA Group (N=23) | Flu mRNA_Ph1_12 YA Group (N=21) | Control Ph1_YA Group (N=23) | Flu mRNA_Ph2_1_YA Group (N=115) | Flu mRNA_Ph2_2_YA Group (N=108) | Flu mRNA_Ph2_3_YA Group (N=137) | Control_Ph2_YA Group (N=120) | Flu mRNA_Ph2_1_Older Adults (OA) Group (N=119) | Flu mRNA_Ph2_2_OA Group (N=122) | Flu mRNA_Ph2_3_OA Group (N=125) | Control_Ph2_OA Group (N=117)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to kidney (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nodular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flu mRNA_Ph1_1 Younger Adults (YA) Group (N=21) | Flu mRNA_Ph1_2 YA Group (N=22) | Flu mRNA_Ph1_3 YA Group (N=23) | Flu mRNA_Ph1_4 YA Group (N=23) | Flu mRNA_Ph1_5 YA Group (N=22) | Flu mRNA_Ph1_6 YA Group (N=25) | Flu mRNA_Ph1_7 YA Group (N=23) | Flu mRNA_Ph1_8 YA Group (N=22) | Flu mRNA_Ph1_9 YA Group (N=23) | Flu mRNA_Ph1_10 YA Group (N=22) | Flu mRNA_Ph1_11 YA Group (N=23) | Flu mRNA_Ph1_12 YA Group (N=21) | Control Ph1_YA Group (N=23) | Flu mRNA_Ph2_1_YA Group (N=115) | Flu mRNA_Ph2_2_YA Group (N=108) | Flu mRNA_Ph2_3_YA Group (N=137) | Control_Ph2_YA Group (N=120) | Flu mRNA_Ph2_1_Older Adults (OA) Group (N=119) | Flu mRNA_Ph2_2_OA Group (N=122) | Flu mRNA_Ph2_3_OA Group (N=125) | Control_Ph2_OA Group (N=117)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 6 (6) | 10 (10) | 8 (8) | 10 (10) | 10 (10) | 14 (14) | 5 (5) | 9 (9) | 8 (8) | 10 (10) | 8 (8) | 11 (11) | 2 (2) | 28 (28) | 41 (41) | 53 (54) | 15 (15) | 20 (20) | 19 (19) | 14 (14) | 10 (10)
Lymphocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal sensation in eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lens disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 2 (3) | 6 (6) | 7 (7) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Oral discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Administration site erythema (General disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 3 (3) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 3 (3) | 2 (2) | 3 (3) | 5 (5) | 8 (8) | 1 (1) | 6 (6) | 7 (8) | 9 (9) | 4 (4)
Administration site pain (General disorders) | 15 (15) | 19 (19) | 21 (21) | 20 (20) | 19 (19) | 22 (22) | 15 (15) | 19 (19) | 18 (18) | 19 (19) | 21 (21) | 18 (18) | 13 (13) | 82 (82) | 86 (86) | 118 (118) | 53 (53) | 63 (63) | 64 (64) | 78 (78) | 41 (41)
Administration site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 3 (3) | 3 (3) | 2 (2) | 3 (3) | 7 (7) | 7 (7) | 1 (1) | 6 (6) | 5 (5) | 8 (8) | 6 (6)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Chills (General disorders) | 4 (4) | 12 (13) | 11 (11) | 14 (14) | 10 (10) | 9 (9) | 15 (15) | 15 (15) | 12 (12) | 12 (12) | 20 (20) | 13 (13) | 0 (0) | 30 (30) | 39 (39) | 73 (73) | 18 (18) | 18 (18) | 19 (19) | 37 (38) | 7 (7)
Exercise tolerance decreased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 10 (10) | 19 (19) | 17 (17) | 18 (18) | 17 (17) | 18 (18) | 16 (16) | 19 (19) | 17 (17) | 16 (16) | 18 (19) | 17 (17) | 9 (9) | 58 (58) | 70 (70) | 103 (104) | 49 (49) | 44 (44) | 51 (51) | 65 (66) | 26 (26)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hangover (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site irritation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site movement impairment (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site paraesthesia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site warmth (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mass (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 2 (2) | 6 (6) | 10 (10) | 4 (4) | 1 (1) | 8 (8) | 5 (5) | 7 (7) | 5 (5) | 9 (9) | 6 (6) | 0 (0) | 5 (5) | 8 (8) | 25 (25) | 2 (2) | 1 (1) | 5 (5) | 14 (14) | 2 (2)
Vaccination site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bronchitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 7 (7) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gonorrhoea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mycoplasma genitalium infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 8 (8) | 7 (7) | 5 (6) | 4 (4) | 3 (3) | 2 (2) | 4 (4)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 4 (4) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Viral rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Avulsion fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibrin D dimer increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 12 (12) | 9 (9) | 10 (10) | 11 (11) | 10 (10) | 9 (9) | 11 (11) | 11 (11) | 7 (7) | 9 (9) | 10 (10) | 0 (0) | 31 (32) | 38 (38) | 48 (48) | 11 (11) | 15 (15) | 27 (30) | 33 (33) | 9 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 5 (5) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Greater trochanteric pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (10) | 21 (22) | 15 (16) | 18 (18) | 15 (15) | 19 (20) | 15 (15) | 16 (16) | 17 (20) | 18 (18) | 21 (22) | 18 (18) | 9 (9) | 57 (58) | 70 (71) | 99 (101) | 35 (36) | 36 (36) | 40 (40) | 57 (58) | 19 (20)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 5 (7) | 7 (7) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 3 (4)
Headache (Nervous system disorders) | 11 (13) | 17 (19) | 15 (16) | 17 (17) | 16 (16) | 17 (22) | 15 (18) | 17 (17) | 14 (16) | 16 (18) | 17 (17) | 13 (13) | 5 (5) | 56 (59) | 59 (63) | 101 (109) | 38 (42) | 39 (40) | 37 (39) | 51 (53) | 20 (20)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paranoia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Poor quality sleep (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 6 (6) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sensitive skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-08-28): https://cdn.clinicaltrials.gov/large-docs/74/NCT05823974/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT05823974/SAP_001.pdf